

| Official Title: | The Implementation of Psychologically Informed Physical Therapy to Prevent Chronification in Service Members With Musculoskeletal Disorders |
|---|---|
| NCT Number: | NCT05132400 |
| Study Number: | s21-01351 |
| Document Type: | Study Protocol and Statistical Analysis Plan |
| Date of the<br>Document: | October 12, 2021 |

# **EIRB Protocol Template (Version 1.4)**

| 1.0 General Information |
|---|
| *Please enter the full title of your study: |
| Factors associated with physical therapy outcomes in active duty service members with musculoskeletal disorders. |
| *Please enter the Protocol Number you would like to use to reference the protocol: |
| PiPT Study * This field allows you to enter an abbreviated version of the Protocol Title to quickly identify this protocol. |
| Is this a multi-site study (i.e. Each site has their own Principal Investigator)? |
| No |
| Does this protocol involve the use of animals? |
| C Yes ⊙ No |
| 2.0 Add Site(s) |
| 2.1 List sites associated with this study: |
| Primary Department Name |
| Navy - Naval Medical Center Portsmouth (NMCP) |
| 3.0 Assign project personnel access to the project |
| 3.1 *Please add a Principal Investigator for the study: |
| Hair, Leslie Chris, DSc CAPT |
| Select if applicable Student Site Chair |
| Resident Fellow |
| 3.2 If applicable, please select the Research Staff personnel: |
| A) Additional Investigators |
| Hope, Timothy Gilman, BS in Biomed. Sciences Associate Investigator Ziemke, Gregg W, CAPT |

| Associate Investigator | | |
|---|---|---|
| B) Research Support Staff | | |
| Stephens, Sam, Psy.D. LCDR<br>Monitor | | |
| 3.3 *Please add a Protocol Contact: | | |
| Hair, Leslie Chris, DSc CAPT | | |
| The Protocol Contact(s) will receive all important system notifications along with the Principal Investigator. (i.e. The protocol contact(s) are typically either the Protocol Coordinator or the Principal Investigator themselves). | | |
| 3.4 If applicable, please select the Designated Site Approval(s): | | |
| Add the name of the individual authorized to approve and sign off on this protocol from your Site (e.g. the Site Chair). | | |
| 4.0 Project Information | | |
| | hie etudy2 | Tf |
| 4.1 * Has another IRB/HRPP reviewed this study or will another IRB/HRPP be reviewing t<br>Yes, answer the questions according to the IRB/HRPP Determination. | ilis study: | |
| | ms study: | • |
| Yes, answer the questions according to the IRB/HRPP Determination. | ms study: | |
| Yes, answer the questions according to the IRB/HRPP Determination. O Yes O No | ins study: | - |
| Yes, answer the questions according to the IRB/HRPP Determination. O Yes O No IRB Name Review Date Determination | ins study: | - |
| Yes, answer the questions according to the IRB/HRPP Determination. O Yes O No IRB Name Review Date Determination No records have been added | ins study: | |
| Yes, answer the questions according to the IRB/HRPP Determination. O Yes O No IRB Name Review Date Determination No records have been added 4.2 * Is this a research study or a Compassionate Use/Emergency Use/HUD project? | ins study: | |
| Yes, answer the questions according to the IRB/HRPP Determination. O Yes No IRB Name | ino study: | |
| Yes, answer the questions according to the IRB/HRPP Determination. O Yes O No IRB Name Review Date Determination No records have been added 4.2 * Is this a research study or a Compassionate Use/Emergency Use/HUD project? O Yes O No 4.3 What type of research is this? | ins study: | |
| Yes, answer the questions according to the IRB/HRPP Determination. O Yes No IRB Name | ino study: | |
| Yes, answer the questions according to the IRB/HRPP Determination. O Yes O No IRB Name Review Date Determination No records have been added 4.2 * Is this a research study or a Compassionate Use/Emergency Use/HUD project? O Yes O No 4.3 What type of research is this? Determination No records have been added | ino study: | |
| Yes, answer the questions according to the IRB/HRPP Determination. O Yes No IRB Name | | |
| Yes, answer the questions according to the IRB/HRPP Determination. O Yes O No IRB Name Review Date Determination No records have been added 4.2 * Is this a research study or a Compassionate Use/Emergency Use/HUD project? O Yes O No 4.3 What type of research is this? Diamedical Research Clinical trial (FDA regulated) Behavioral Research Educational Research Psychosocial Research Oral History | | |
| Yes, answer the questions according to the IRB/HRPP Determination. O Yes O No IRB Name Review Date Determination No records have been added 4.2 * Is this a research study or a Compassionate Use/Emergency Use/HUD project? O Yes O No 4.3 What type of research is this? Biomedical Research Clinical trial (FDA regulated) Behavioral Research Educational Research Psychosocial Research Oral History Other | | |

| uses, studies, or a | nalyzes the informat | tion or biospecimens; or | or interaction with the individual, an |
|---|---|---|---|
| ⊙ Yes C No | | | |
| .7 * Do you believe t | his human subjects | research is exempt from | IRB review? |
| O Yes 🖸 No | | | |
| .0 Personnel De | | out EIRB access that are | e not previously entered in the protoco |
| Name:<br>(Last, First, M.I.)<br>Campello, Marco | Phone Number: | Email Address: | Associated<br>Institution: |
| Role on Protocol: | 212-255-6690 | marco.<br>campello@nyulangone.<br>org | New York<br>University |
| Name:<br>(Last, First, M.I.)<br>Weiser, Sherri | Phone Number: | Email Address: | Associated<br>Institution: |
| Role on Protocol: | 212-255-6690 | sherri.weiser-<br>horwitz@nyulangone.<br>org | New York<br>University |
| Name:<br>(Last, First, M.I.)<br>Oh, Cheongeun | Phone Number: | Email Address: | Associated<br>Institution: |
| Role on Protocol: | 212-263-3394 | ohc03@nyumc.org | New York<br>University |
| Name:<br>(Last, First, M.I.) | Phone Number: | Email Address: | Associated<br>Institution: |
| Mowery, Hope C. Role on Protocol: | 212-255-6690 | Hope.<br>Mowery@nyulangone.<br>org | New York<br>University |
| AI | | | |

| <ul><li>Yes</li><li>No</li><li>N/A</li></ul> | | | |
|---|---|---|---|
| Research Monitor Qualification Ensure the individual has expert study and is independent of the | ise consistent with the nature of | f risk(s) identified within your | |
| Research Monitor Role: | | | |
| We have identified a clinical psyc<br>Research Monitor. | chologist at NMCP, LCDR Sam St | tephens, to serve as our | |
| A primary focus of our study is the outcomes. Our participants will a participation in this study will not us in navigating any emotional dunexpected problems that may expected problems. | Iready be receiving treatment b<br>t alter their course of treatment<br>istress-related adverse events, | y a physical therapist, and<br>. Our research monitor will as | |
| If applicable, you may nominate | an individual to serve as the Re | esearch Monitor: | |
| Selected Users | | | |
| Sam Stephens, Psy.D. | | | |
| 6.0 Data/Specimens 6.1 Does the study involve the subjects)? | e use of existing data or spe | cimens only (no interactio | n with human |
| C Yes ⊙ No | | | |
| 7.0<br>Funding and Disclo | osures | | |
| 7.1 Source of Funding: | | | |
| | Funding Type | Amount | |
| 7.1 Source of Funding: Funding Source Congressionally Directed Medical Research Program (CDMRP) | Research Development : Testing and Evaluation (RDT&E) funds | Amount 1527509 | |
| Funding Source Congressionally Directed Medical Research Program | Research Development : Testing and Evaluation (RDT&E) | | |
| Congressionally Directed Medical Research Program (CDMRP) | Research Development : Testing and Evaluation (RDT&E) | | |
| Congressionally Directed Medical Research Program (CDMRP) | Research Development : Testing and Evaluation (RDT&E) funds | of a personal interest or f | |

If Yes, complete and attach Conflict of Interest forms for all key personnel

## 9.2 Background and Significance:

Include a literature review that describes in detail the rationale for conducting the study. Include descriptions of any preliminary studies and findings that led to the development of the protocol. The background section should clearly support the choice of study variables and explain the basis for the research questions and/or study hypotheses. This section establishes the relevance of the study and explains the applicability of its findings

Chronic pain from Musculoskeletal Disorders (MSD) poses a significant problem for Active Duty Service Members (ADSM) and are the main reason for separation and long-term disability. <sup>1-4</sup> Overseas conflicts in the last decade have contributed to a rise in reported MSD among ADSM. <sup>5</sup> Sailors and Marines who experience MSD have the highest level of attrition from these disorders among all military branches. <sup>6-8</sup> In a study conducted on two deployed United States Navy aircraft carriers, Hebert et al. (2004) <sup>9</sup> found that MSD comprised 40% to 43% of all sick call visits during deployment. Lewis Shattuck et al. (2016) <sup>10</sup> found that 57.7% of ADSM aboard a Navy carrier reported MSD symptoms over the course of one year; twenty percent of whom had symptoms that interfered with their daily activities on board ship. The current investigators studied all Navy ADSM and found that the rate of conversion from first career limited duty assignments to the fitness for duty assessment or physical evaluation boards (PEB) was 15% for MSD cases. Only 28% of those referred to PEB return to full duty. <sup>11,12</sup> It is apparent that MSD deserve our attention. Despite this, there is little research into effective treatment approaches for MSD in Navy ADSM.

#### Risk factors associated with MSD-related disability in ADSM

Several factors have been shown to be strongly associated with disability from MSD. Studies looking at work outcomes in military populations emphasize a biopsychosocial perspective that includes a variety of factors. Feuerstein et al. (1997)<sup>13</sup> and Berkowitz (1999)<sup>14</sup> identified characteristics associated with disability in ADSM including younger age, lower rank, poor aerobic conditioning, high work stress, worries and low social support. Lincoln et al. (2002)<sup>15</sup> also found similar factors to be associated with disability from MSD in ADSM such as pay grade, diagnosis, length of service, age, military occupational specialty, job satisfaction, previous history of MSD, smoking, work stress and job demands. Schoenfeld et al. (2014)<sup>16</sup> found that MSD, psychiatric conditions, and lower rank accounted for 78% of the variance in unfavorable Physical Evaluation Board (PEB) outcomes in soldiers with a variety of health complaints.

Studies specific to Navy ADSM are few but echo some findings from studies of other military branches. Stephanie Booth-Kewley et al. (2009)<sup>17</sup> explored a variety of psychosocial factors contributing to attrition from basic training due to MSD in Marine Corps recruits but found only expectations about graduation and career intentions to be predictive in the final regression analysis. In a later study, the same researchers found similar results in a

one-year follow-up of injured marines. Individuals who had high recovery expectations at baseline were over five times as likely to be recovered at follow-up as individuals who had low expectations (OR = 5.18,  $p \le .01$ ). <sup>18</sup> A longitudinal study conducted by the present investigators examined the relationship between known modifiable psychological risk factors and work outcomes among ADSM who were not deployed and found that fear of activity was predictive of work status twelve weeks after a reported back injury. <sup>19</sup> Taken together, these studies provide clear scientific evidence linking psychosocial factors with increased risk of disability following MSD in ADSM and support additional investigation into Navy members.

The biopsychosocial model of pain and disability explains the multidimensional nature of MSD. This model emphasizes the interplay of physiological and psychological (cognitive, affective, and behavioral) responses to pain and how they interact with the social environment to ameliorate or maintain pain and dysfunction. For example, when there is prolonged pain, cortical changes result in altered muscle response patterns such as abnormal dynamic muscle control. <sup>20,21</sup> In addition, stress hormones that accompany these painful conditions enhance pain transmission. <sup>22</sup> These changes result in cognitive appraisals of pain as unremitting and individuals often express anxiety about their future and suffer depression from feelings of helplessness and hopelessness. Many develop a fear of movement that is reflected in the social dimension as restriction of work and social activities. <sup>23</sup> This pattern decreases the likelihood of recovery as it is self-sustaining.

This model is applied to clinical practice by identifying various elements as risk factor categories, or 'flags'.<sup>24</sup> Red flags are clinical indicators of serious underlying conditions that warrant further medical intervention such as the presence of systemic diseases. Orange flags can be considered the psychiatric equivalent of red flags and include serious psychiatric pathology that may interfere with recovery such as clinical depression and Post-traumatic Stress Disorder (PTSD).<sup>25</sup> Yellow flags are modifiable psychological or behavioral risk factors associated with unfavorable clinical outcomes. Common yellow flags are negative beliefs about recovery, feelings of distress and inability to cope with pain. Blue flags are the workers' perceptions of the work environment such as perceived work stress or lack of social support. Black flags are characteristics of the system or the environment in which a person functions such as the nature of the work or the insurance and compensation system of the workplace.<sup>25</sup> Recently pink flags, which are protective from poor outcome such as self-efficacy and positive outcome expectations, have also been identified and should be considered when assessing risk.<sup>26</sup>

# Evidence of effectiveness of Cognitive Behavioral Therapy (CBT) in modifying psychological risk factors

Yellow flags are considered modifiable through clinical intervention. CBT, derived from a well-established mode of psychotherapy, has been developed to address modifiable psychological risk factors for chronicity and poor outcome in patients with MSD. <sup>27-30</sup> CBT is rooted in the work of Aron Beck, who identified automatic thoughts or responses to stimuli that result in affective states that may interfere with adaptive behaviors and proposed techniques to alter these thoughts. <sup>31</sup> The emphasis on modifiable factors is of critical importance to the development of effective interventions for treating MSD. It has been shown that there is a clear relationship between the presence of modifiable yellow flags and future clinical and occupational outcomes. Indeed, factors such as fear-avoidance beliefs, distress, somatization, and pain catastrophizing are associated with high risk of a poor outcome such as chronicity in patients with low back pain (LBP). <sup>26,30,32-34</sup>

Using CBT to target yellow flags, especially when they are at high levels, leads to more positive outcomes. <sup>25,35,36</sup> Systematic reviews show moderate evidence that treatments that address psychological factors using cognitive-behavioral techniques in conjunction with PT are effective in reducing symptoms and limiting disability among individuals with sub-acute MSD. <sup>37-39</sup> A recent study showed CBT to be cost-effective in treating chronic pain. <sup>40</sup> Furthermore, it has been shown that patients with psychological risk factors do not benefit from a biomedical approach alone but do benefit from a combined approach. <sup>36,39,41,42</sup> For example, patients with Low Back Pain (LBP) who express fear of activity can be treated successfully only when these fears are addressed. <sup>30</sup>

#### Benefits of Psychologically-informed Physical Therapy (PiPT)

Identification and modification of yellow flags has been shown to be effective in reducing or preventing chronic or recurrent disability in patients with MSD. 36,41,43,44 Recently, it has been proposed that this should be done by physical therapists who have early and prolonged access to patients. Other advantages of having physical therapists address yellow flags are that CBT administered by a psychologist is expensive, may not be readily available and patients may be reluctant to seek psychotherapy due to stigma.

PiPT, sometimes called psychologically based PT, is an approach designed to incorporate the concepts of CBT for pain management into routine clinical PT practice in order to modify maladaptive responses associated with chronicity. The goal of PiPT is to promote a fast and optimal recovery by removing psychological obstacles, obviating the need for referral to a psychologist and facilitating triage to other health professionals in a timely manner when needed. PiPT training includes education about the neuropsychology of pain, patient communication skills, and identification of psychosocial risk factors for chronicity and treatment approaches that include reassurance, relaxation, and psycho-behavioral reactivation. Currently, PT training is based in the biomedical model, which posits a direct relationship between the nature and severity of the injury and the symptoms reported by the patient. In this model, the objective of treatment is to address the physical cause of pain or disability in an effort to improve outcomes without taking into account the psychosocial nature of the risk factors for chronicity and disability. A shift in treatment from the biomedical paradigm to a biopsychosocial paradigm requires education and training.

Studies have found that physical therapists who acknowledge the importance of addressing psychological risk factors in patient care often feel ill equipped to do so. 46,47 There is a growing body of literature suggesting that physical therapists have the potential to assimilate

biopsychosocial principles into their traditional biomedical training. $^{48-51}$  However, it is yet unknown how well such training translates into clinical application. Studies exploring the impact of this training on patient outcomes are promising but are limited by small sample sizes or low response rates. $^{52-54}$ 

In one recent larger study, Overmeer et al developed an eight-day training course for physical therapists in PiPT including questionnaire administration, the biopsychosocial model, yellow flags, behavioral principles, communication, addressing fear of movement, and role playing.<sup>45</sup> In a randomized clinical trial (RCT) examining the effectiveness of this training, the investigators found that while attitudes and knowledge of the physical therapists shifted in the expected direction, their behavior did not. Furthermore, training did not improve patient outcomes. However, patients with high of levels catastrophizing and depression showed better outcome regarding disability when the attitudes of therapists changed from purely biomedical to psychologically-based.<sup>55</sup> The authors point out that a one-time course is insufficient for changing behaviors, even if attitudes are altered. Ongoing education and reinforcement is needed. This sentiment is echoed in a study by Nielsen et al. (2014)<sup>49</sup>, where trained physical therapists stated a preference for more role-play experience prior to implementing treatment. Secondly, Overmeer et al.  $(2011)^{55}$  speculate that their topics were too broad and did not focus on specific ways to address yellow flags. Finally, they posit a possible selection bias in that participants were interested in learning about yellow flags, so they may have already been exhibiting different behaviors than other physical therapists.

Our research group has experience in training Navy personnel to address psychological risk factors. We designed an education and training program for an interdisciplinary team at the Navy Medical Center Portsmouth (NMCP). Team members were trained in the biopsychosocial model as a group and then individually by experts in their field. The purpose of this training was to teach physical therapists, psychologists, and physicians how to work in an interdisciplinary team. In a pilot randomized controlled trial, we tested the feasibility of implementing an interdisciplinary work restoration program based on this training called "Backs to Work" in a Navy and Marine Corps setting for ADSM with work-limiting low back pain. We found preliminary evidence that those randomized to CBT and PT had improved perception of function as compared to usual care and there was a trend of decreased fear of activity and pain catastrophizing in the intervention group as compared to usual care. Se

Furthermore, we developed a PiPT course to train PT personnel aboard an aircraft carrier in a case-controlled cohort pilot study comparing PiPT to usual care. Results demonstrated the feasibility of implementing this intervention onboard US Navy aircraft carriers. <sup>57</sup> Trained PT personnel achieved a priori criteria for feasibility by obtaining passing knowledge scores following training, completing clinical notes indicating PiPT implementation and participating in regular case reviews in which they discussed their treatment plans via phone conference with the research team. Feedback from the PT staff who stated that their treatment paradigm and practice had changed from a biomedical to a biopsychosocial model after training also confirms successful transfer of PiPT training into clinical practice.

We found evidence for the effectiveness of PiPT in the carrier study as well. Subjects in the intervention arm reported learning coping strategies that are associated with good outcomes. Responses to the question "Please list the most important things you learned in physical therapy?" differed between the two groups. Among subjects on the intervention carrier, 33.7% indicated they had learned concepts consistent with PiPT treatment based on a priori analysis criteria developed by the investigators. For example, one intervention subject said, "Stress and physical pain have a connection". In contrast, none of the subjects from the control carrier responded in this manner. <sup>11</sup> Our experience with PiPT training has informed the development of the present proposal.

In our interdisciplinary training for the RCT described above, we avoided some of the weaknesses highlighted in previous studies by giving specific examples of how to implement guideline-based care for each discipline and by providing weekly teleconferences to answer questions, discuss difficult cases and reinforce training. <sup>56</sup> In addition, we encouraged the use of self-care techniques to reduce patient reliance on health care professionals. This further distinguished our approach from Overmeer's. In our training for US Navy PT staff aboard a carrier we replicated our original training while incorporating important aspects found to be effective in other studies, such as ongoing role-playing and case-examples once the PT staff was deployed through teleconference. <sup>57</sup>

The long-term objective of our research is to implement PiPT in different settings and for different cohorts of patients with MSD, throughout the Military. Therefore, we propose a full-scale study replicating the design and methods used in our pilot carrier study to test the feasibility and short- and long-term effectiveness of PiPT on psychological and functional outcomes in ADSM seeking care for MSD at a shore based rehabilitation setting; Navy Medical

Center Portsmouth (NMCP). ADSM who seek care for MSD at NMCP may differ from patients aboard a carrier in terms of type and duration of MSD, rank, deployment status and environment. For example, most of the MSD on the carrier were acute and unlikely to be severe. The NMCP sees all ADSM with MSD regardless of severity and duration. Therefore, we wish to establish feasibility and effectiveness of PiPT in this setting to augment the generalizability of our findings. The results of this study along with those from the carrier study will allow us to modify our rehabilitation strategy to address the needs of specific Navy cohorts across different phases of care in different health care settings. The ultimate goal is to decrease MSD-related chronicity leading to disability in ADSM in support of combat readiness.

# 9.3 Objectives/Specific Aims/Research Questions:

Describe the purpose and objective(s) of the study, specific aims, and/or research questions /hypotheses

Our study objective is to establish the feasibility of implementing a psychologically informed rehabilitation strategy while concurrently assessing its' effectiveness in ADSM with MSD seeking care in a US Navy shore-based health care setting. This intervention is intended to improve the management of chronic pain in order to optimize ADSM function.

# Specific aims

- 1. Demonstrate the feasibility of implementing PiPT in a US Navy shore-based health care setting. We will analyze SOAP notes to assess whether the clinicians have applied aspects of the training in the treatment given to the patients and they are reflected in the notes.
- 2. Document and compare baseline risk factors related to pain interference in two cohorts of patients with MSD.
- 3. Demonstrate the effectiveness of a PiPT intervention on psychological and functional work outcomes in a comparative effectiveness trial through a relative increase in protective follow-up measures such as quality of life, self-efficacy, and satisfaction and a relative decrease in detrimental measures like pain catastrophizing, fear of movement, and distress.

# 9.4 Study Design:

Describe study design in one to two sentences (e.g., prospective, use of existing records/data /specimens, observational, cross-sectional, interventional, randomized, placebo-controlled, cohort, etc.). Specify the phase – Phase I, II, III, or IV – for FDA-regulated investigational drug research

We are proposing an observational prospective comparative cohort study. This study meets the criteria for a hybrid type 3 study; a hybrid type 3 study tests an implementation/strategy while observing/gathering information on the clinical intervention and related outcomes.<sup>58</sup>

# 9.5 Target Population:

Describe the population to whom the study findings will be generalized

Active duty service members receiving physical therapy for musculoskeletal disorders.

#### 9.6 Benefit to the DoD:

State how this study will impact or be of benefit to the Department of Defense

This study will demonstrate the feasibility and efficacy of implementing PiPT training at a military treatment facility in improving outcomes of musculoskeletal disorders. The ultimate goal is to decrease MSD-related chronicity leading to separation and disability in ADSM in support of combat readiness.

## 10.0

# Study Procedures, Data Management, and Privacy

### 10.1 Study Procedures:

Describe step-by-step how the study will be conducted from beginning to end

#### Phase I

## Recruitment and Consenting

- Research staff will review the PT clinic's schedule for patients scheduled for initial
  evaluation, then request an introduction from the therapist if appropriate (patient must
  be scheduled for at least 4 physical therapy sessions).
- Research staff will brief the patient on the study.
- If the patient is interested, the researcher will show them to the private study room, screen them for eligibility, and then ask them to review the consent form. The researcher will remain in the room to answer any questions.

# Treatment

- After signing the consent form, the participant will complete a paper form collecting contact information for follow-up and demographic information. At this point, the participant will be assigned a participant ID number. The researcher will verify the participant's diagnostic code and therapist using AHLTA afterward.
- Before the participant's next PT appointment, the participant will complete the baseline
  questionnaire battery, a 139 question survey battery. The participant may complete the
  battery immediately on paper, or at a later date online using a link to REDCap that will be
  sent via encrypted email. This battery must be completed before their next appointment.
- Participants will receive standard PT care as prescribed and scheduled by their therapist.
   Participation in the study will not alter their care plan.
- Participants will complete follow up questionnaire batteries after their 4<sup>th</sup> PT appointment\*, 6mo and 12mo post enrollment. The first follow-up questionnaire is a 77 question survey battery. The second and third follow-up points use a 68 question battery. All follow-up questionnaires will be completed remotely via REDCap.
- We will collect de-identified SOAP notes from randomly selected participants and review
  them for verbiage indicating that the therapist employed principles of PiPT. We will collect
  up to 30 SOAP notes, pertaining to various physical therapists and throughout various
  stages of treatment.

## PT Training

Following the completion of Phase I recruitment, PT staff will be trained in PiPT by the NYU personnel. NYU personnel intend to deliver the training in person; however, they are prepared to deliver virtual, real-time training should COVID protocols make face-to-face training unfeasible.

- PT staff will receive a knowledge quiz at the end of their training sessions to document successful completion of training. PT staff must obtain a passing score (85% or above) on this quiz to be considered proficient.
- We will also assess the PT staff's confidence in implementing PiPT using a seven point Likert scale self-rating derived from a previous study.
- Furthermore, staff will be evaluated on the accurate identification and management of yellow flags using case studies.
- Once the staff shows proficiency in delivering PiPT, the second study phase will begin.
   There will likely be some overlap between the follow-up data collection of Phase I and the training period.
- After initial training and as Phase II recruitment begins, staff will receive weekly reinforcement sessions for one month, after which they will receive further reinforcement sessions on a biweekly basis as needed.

During training, PT staff will be asked whether they have had previous experience with PiPT. If so, participants who saw these providers, whether during Phase 1 or 2, will be analyzed for a possible confounding effect.

#### Phase II

#### Recruitment and Consenting

- Recruitment for Phase II will largely proceed as with Phase I (pending unforeseen changes in the PT department's process). The only major change is that when researchers screen the schedule for evaluation appointments, they will also verify that the corresponding therapist completed the PiPT training.
- Research staff will brief the patient on the study.
- If the patient is interested, the researcher will show them to the private study room, screen them for eligibility, and then ask them to review the consent form. The researcher will remain in the room to answer any questions.

#### Treatment

- After signing the consent form, the participant will complete a paper form collecting contact information for follow-up and demographic information. At this point, the participant will be assigned a participant ID number. The researcher will verify the participant's diagnostic code and therapist using AHLTA afterward.
- Before the participant's next PT appointment, the participant will complete the baseline
  questionnaire battery, a 139 question survey battery. The participant may complete the
  battery immediately on paper, or at a later date online using a link to REDCap that will be
  sent via encrypted email. This battery must be completed before their next appointment.
- Participants will receive PT care as prescribed and scheduled by their therapist.
   Participation in the study will not directly alter their care plan.
  - During Phase II, we anticipate that therapists who completed PiPT training will
    incorporate the training into their standard care. We will not ask therapists to give
    differential treatment to patients who are enrolled in the study.
- Participants will complete follow up questionnaire battery after their 4<sup>th</sup> PT appointment, 6mo and 12mo post enrollment. The first follow-up questionnaire is a 77 question survey battery. The second and third follow-up points use a 68 question battery. All follow-up questionnaires will be completed remotely via REDCap.
- We will collect de-identified SOAP notes from randomly selected participants and review them for verbiage indicating that the therapist employed principles of PiPT. We will collect up to 30 SOAP notes, pertaining to various physical therapists and throughout various stages of treatment.

We chose to conduct this study in sequential cohorts rather than conducting the two cohorts (PiPT and non-PiPT) in parallel because there are no comparable sites with similar characteristics such as type of subjects, catchment area size and availability of the health care team in the Navy.

\*We chose the 4th visit as the first follow-up point for two reasons. First, we expect to see a difference between groups on study outcomes at that point. Secondly, since according to the former head of the NMCP department of physical therapy (PI) the average number of visits at the outpatient PT clinic is 6, the 4th visit will allows us to capture complete data.

#### 10.2 Data Collection:

Describe all the data variables, information to be collected, the source of the data, and how the data will be operationally measured.

# Intake Form (Demographics) C o V VII aR C A e rie i R C T as t I OD a A OD o t B P L T s L o ye i ps n e t

```
I DF
n Sier
Gtnme
e agloen
n keg R/
de Itrea
e Feas
rompp
r hio
m cn
                            s s
                                    e
e
Dr
n Sime
t no Rn
ge Rn
ge Itap
o mhin
m se
FF
MI
DF
Dr
an Sime
rit no R
taglgen
alkersa
ate Itap
to mhin
sm cs
                           D
I D
I e
Simy
t no e n
k e r /
cie Ita /
t e p
y o mhi
r c
m s
          Ι
                           D
I D
I e S
n Simel
R a glg ctn
a k e r fr/
c e Ita o a
e F e p m
o mhiLi
r c st
s
           Ι
e DF
g I e e
t t no R
haglg e /
of k e r s a
r e p o
m n
```

his D T e Sim n o R k glg e s/ e r a a a a o a o a o a o a mhi С S S D Da e t aln Sime u t no( ti k glg d n erd/ n F Do e p O mhiN t m s y ) D m st A o n Hg Lr Ta a Ap ; hi Fi c t S D e C m<sub>D</sub> Ао . g 1 n L r 1 , Та Ар hi d

Evaluation Date: Because participants will be consented and fill out the intake form on the day of their PT evaluation, the research staff member will simply record the current date that the form is completed.

We will require a DSA to harvest those last two variables.

# Questionnaires/Outcomes

The self-report questionnaire batteries are largely composed of the validated survey tools and single-item questions.

- 1. The Pain Disability Index (PDI) will measure pain interference. <sup>60</sup>
- 2. Catastrophizing will be assessed by the Pain Catastrophizing Scale (PCS). 61
- 3. Fear avoidance beliefs will be assessed using the Fear Avoidance Beliefs Questionnaire (FABQ). 62,63 (Excluding "I have a claim for compensation for my pain," no relevance).
- 4. Psychological distress will be measured using the Hospital Anxiety and Depression Scale (HADS). 64-66
- 5. Self-efficacy will be assessed using the Pain Self-Efficacy Questionnaire (PSEQ).  $^{67-70}$
- Positive outcome expectations will be assessed using a 5 point single item scale developed for the military population by Stephanie Booth-Kewley et al. (2009).

- 7. Satisfaction with process of care will be measured by the "process of care" subscale of The MedRisk Instrument for Measuring Patient Satisfaction (MRPS). 71,72
- 8. Outcome satisfaction (single item scale): 'If you had to spend the rest of your life with the symptoms you have right now, how would you feel about it? This is derived from the Core Outcome Measures Index (COMI) questionnaire.<sup>73</sup>
- 9. Clinical Depression: The Center for Epidemiologic Studies Depression Scale (CES-D).  $^{74,75}$
- 10. Anxiety Disorder: General Anxiety Disorder Screener (GAD-7). 76
- Post-Traumatic Stress Disorder (PTSD) will be assessed using the PTSD Checklist Military version (PCL-M).<sup>77,78</sup>
- 12. Job satisfaction (single item scale): "Taking everything into consideration, how do you feel about your job as a whole?" taken from Dolbier et al. (2005): <sup>79</sup>
- 13. Work stress (single item scale): "Taking everything into consideration, how stressful is your job as a whole?"
- Organizational commitment (single item scale): Commitment will be assessed by the affective dimension of the Commitment Scale. 80-83
- Job social support: Subject's relationships with co-workers and social environment at their job, drawn from the Deployment Risk and Resilience Inventory-2 (DRRI) unit support subscale.<sup>84</sup>

Injury history: affected body part(terminology adopted from Barrel matrix.<sup>85</sup>), time since onset, other MSD comorbidities, episode recurrence, previous MSD and pain intensity. Baseline Questionnaire Battery

- 139 questions charted below and one open field question on any barriers to treatment the participant perceives.

```
C
o
   V
Ш
s_T C S
e o el
li n e
li r foctn
n foctn
e u fr/
 e u fr/
  e
It
d m
r e Li
v m = =
v rst
   D
   e S
e Simel
linoe
nglg ctn
eerfr/
SItaoa
uepm
r mhiLi
   c st
В
a
```

```
P li
ri n
m e
ae

rueS

yrSimel

Iynoe

njeglgct

uyerfr8

r, Itao5

yFepm

LomhiLi

oll cst

cos

aw

ti-

oU
         р
1
         2
        3
                                >
                                4
                                W
                                e
                                e
                                k
                                s,
        В
B S,
Tia D 4
ms e 4
e e Sim 1
si li n o 2
n n glg w n
c e e r e /
e SIta e
o u e p k
n r mhi
s v c s,
ete s 
y 1
                                1
                                2
                                W
                                e
e
                                k
                                s
E
piB
sa D
os e
deSim
elinoe
Rnglgsn
eeer/
cSItaN
uuepo
rrrmhi
ev c
ne s
cy
e
B
P a D r s T e Y e m e li o
```

```
vinogsn
o e Itr / /
 u Se a N a
sumpo
Mrhi
Svc
 Dе
             s
     У
     В
      a
      s
      е
     li
     n
     e
     S
    u D
Preo
aiv Sim-
neno-
iny glgon
t, ers/
e F Itaca
noepal
sill mhie
     w s
     U
     p
     1
     2
     3
3
B
Ma D
S s e S
D e Simel
c li n o e
o n glg ct 8
me e r fr 5
o u e p m
r r mhiLi
bi v c st
ty
B
     В
     S
    e
   li I
On n
ue d
tcS e
ou p
mr Sie 0
e vnn -
e e gld 5
x y e e s 7
p , it n c
e F e t al
ctomV e
a ll a
ti o ri
o w a
n - bl
               e
```

```
U
  1
  В
  a
  s
  e
 li
 n
 e D
 s e
Seuprescondingers e
    bl
 U e
 p
  1
  2
 3
  В
  a
  s
  e
 li
      0
 n
U en
     S
 p
  1
 2
 3
  В
  a
  S
  е
 li
 n
     0
 e
 S D-
 u e6
 r ps
    e c
n
d
```

```
efe P e al 6 fi y S n e 7 c , E t ; a F Q V 1 c o a 0 y ll riq
    o au
    w ble
           e st
    U
            io
             n
    р
    1
              S
    2
    3
    В
     a
    S
    e
    li
 n
 Pe D-
aiS e4
aiS e 4
nu ps
Cr e c
a v nal
t e de
a yPe; 6
st, Cn 1 1
r FSt 3
o o Vq
p II a u
hio rie
ziw a st
n - blio
g U e n
p s
    p
            S
    1
    2
    3
    В
    a
    S
    е
    li
    n
            0
  e D-
e D-
FS e 6
e u ps
ar e c
r v n al
ofe d e
my A e; 6
o, B t 5
e o V q
mll a u
 eorie
nwast
          a st
           blio
    Uen
    p
            S
    1
    2
```

```
В
     e
    li
               4
    n
    e Dp
    s et
    u ps
u ps
r ec
D v nal
is y H e;
tr y A n 1
e F S V q
s II a u
o rie
                     6
4
     w ast
            blio
    Uen
                 s
    p
     1
     2
     3
        Α
        ff
                 5
e p
Bct t
r se C k
c li o n rt
m emu 4 0
it umd u
e vn r st
t ys
        e
                io
    y s
C
                n
                S
         al
         e
                 5
                p
t
JB t
oa Li
bs Ck
se oe
oli nrt
cinR u 1
s SR n 2
u u dq
pr eu
pv re
oe st
rty io
                     8
4
                 n
                 s
                 1
                -
5
s
c
    В
    a
s
e
            C
0
```

```
P li P n al
T n C foe 7
S e L u; 7
S - n 1
u M d 7
               e q
              r u
      ٧
      e
                   e
                   st
                   io
                   n
                   s
                   0
                   -
                   3
     В
                   S
    a
a s
Ds Cc
ee oal
pliCne
rnEfo; 7
eeSu24
siuDdq
or eu
nv re
                   st
      е
                   io
                   n
                   s
                   0
                   3
      В
a 3
s C c
e o al
A li G n e
n n A fo; 7
xi e D u 7 6
tyu 7 d q
r e e
      a
                   e
             r
                   st
      е
                   io
                   n
                   s
      В
      a
      li
      n
MS
eu

trTOY
Hyerfos/
alerfos/
toen
al'Fitd
o
Co
aw
e
aw
e-
aw
e-
e
       e
      u
     р
1
```

```
3
    В
 J a
Ja
os C
beSio 1
s linn-
anglfo5
tieeus 9
sfSitnc
auedal
ctrmee
iov r
ne
  У
    В
  a
 Ws C
ws C
o e Sio 1
r li n n -
k nglfo5 n
stee u s /
r Sit n c a
euedal
srmee
svr
    e
    У
                F
                ul
                В
                D
     a
                u
     s
                t
     e
                У
     li
     n
                Li
     e
                m
    S
                it
u it
u e
Dr Cd
u v Sio D
tyen n u
S y glfot n
t , e u y ,
a Fit n ,
u ll me
s o r
    u
 so r
                d
     W
                В
                0
     u
                a
     p
                r
     1
                d
     2
                O
    3
                t
                h
                e
                r
P
e D
eiB e F
va pr
es e e
d e Sin e
b lind R
angle e
rree n
```

```
ieSItt s 1
    rsue V p 1
             r ma o
                                  ri n
   о е
                                  a s
                                  ble
   Follow-up Questionnaire Batteries
                                                       Post 4<sup>th</sup> treatment session- 77 items long, including one open field question
                                                       6 and 12mo - 68 items (excludes MRPS scale and outcome expectation)
               C
               0
                  o
                                      p s
               n
               t
               В
               a
               S
             е
  P li
  ri n
  me
  a S
ru D
yr e S
IvSimel
  nenoe
j yglg ct
u , e r fr
r FIta o
 y o e p m
L ll mhiLi
 oo cst
cws
a-
tiU
   ор
   n 1
               2
               3
               В
               а
               S
               S
Preadored Preado
```

```
sill Ithial
        toece
       y wms
                          U
                         p
                         1
                         2
                         3
                          В
                         a
                         S
                   e I
     Olin
und
     tce e
   oS p
muSie0
ernn-
evgld 5
xeees 7
pyitnc
e, et al
   ao a
till ri
     oo a
nw bl
                                                           е
                       U
                       p
                         1
                          В
                          a
                          S
                          е
                       li
                       n
                         e D
                         S e
                       и р
 Qrepored Processing Pr
     of ne val
Lill mae
fe ri
                          w a
                                                         bl
                         U e
                         p
                          1
                         2
                         3
                          В
                          a
                          S
                         е
                       li
                                                                0
                     n
 pe D-
ai p0
```

```
nr es
I v nc
ne dal
t yPee
e, Dn; 0
rfFI t 7
eo Vq
r II a u
eo rie
n w a st
c - blio
e U e n
     р
               S
     1
     2
     3
      В
      a
      S
      e
     li
                    0
     n
     e D-
     S e 6
     u ps
u ps
Srecelv nal
f-epde
efyse; 6
fi, En 17
cFQtO
ao Vq
cll au
     W
              a st
              blio
     Uen
                S
     p
     1
     2
     3
     В
     a
     S
      е
     li
n 0
Pe D-
aiS e 4
nu ps
Cr ec
a v nal
te de
a yPe; 6
st, Cn 1 1
r FSt 3
o o Vq
pll a u
hio rie
ziw a st
n - blio
g U e n
p s
     1
```

```
,
3
B
    a
    S
    e
    li
    n
             0
    e D-
FS e 6
e u ps
ar e c
r v nal
ofe d e
my A e;
o, B t 5
e o V q
mll a u
e o rie
n w a st
t - blio
                  6
2
    U
         e n
    p
    2
    3
    В
    а
    S
    е
    li
               4
    n
    e
         Dρ
          e t
    S
          p s
    u
u ps
r ec
v nal
ise H e;
tr A n 1 4
s o V q
s II a u
o rie
w a st
           blio
    U
         e n
               s
    1
    2
    ,
3
B
    a
    S
    e
    li
    n
```

```
alFen/n
  t o Itd N/
 h II e e o a
 Comr
aw
r -
e u
       p
       1
      2
      3
S
a D
ti e 5
a F e k
ioll Ede; 7
it - Sf e K
ioll Ede; 7
it - St e k
ioll Ede; 7
it - I t q
p p K a io
p p K a io
e e s
S D e e s
sfo C p
a ll O M n b f
c to M n c
u 2 e ri
t c, ma
o 3
m
                        F
                       ul
                       1
       В
                        D
       a
                       u
       s
                        t
       е
                       y
;
       li
       n
                       Li
       e
                        m
S m
S it
D r C d
t v Sio D
y y glfo t /
S , e u y a
a o e d M
u o r d
s w B
       S
                       e
d
B
```

1 d 2  $\cap$ t h е D p lell e a o Sin wn d n - gle e u e n d p Itt fr 1 e V o , ma m2 ri a s h 3 bl<sup>e</sup> SOAP Note Review Researchers will review the randomly selected, de-identified SOAP notes for verbiage indicating that the therapists identified and applied principles of PiPT, such as references to yellow flags like fear avoidance behavior. These SOAP notes and their reviews will not be assigned a Subject ID number or otherwise be associated with their corresponding demographic information or questionnaire responses.

10.3 At any point in the study, will you request, use, or access health information in any form, including verbal, hard copy and electronic?

10.4 Review the definitions below and respond to the following two questions. If you are not sure of the answers, email DHA.PrivacyBoard@mail.mil for assistance. The Military Health System (MHS) is defined as all DoD health plans and DoD health care providers that are organized under the management authority of, or in the case of covered individual providers, assigned to or employed by, the Defense Health Agency (DHA), the Army, the Navy, or the Air Force MHS workforce members are employees, volunteers, trainees, and other persons whose conduct, in the performance of work for the MHS, is under the direct control of the MHS, whether or not they are paid by the MHS. MHS business associates are persons or entities that provide a service to the MHS and require protected health information (PHI) to provide the service.

# Are you an MHS workforce member?

Yes, I am an MHS workforce member

O No, I am not an MHS workforce member

#### Are you an MHS business associate?

C Yes, I am an MHS business associate

| O No, I am not an MHS business associate | |
|---|---|
| 10.5 Have you consulted with an MHS data expert to determine the data elements required for your study? | |
| Consulting with a data expert often saves time la expert can advise on the data available in the number that data and the methods for encrypting and col MHS data expert, send an email to: (DHA.Privacon Yes, then complete the questions below accord No, then complete the questions below accord | merous MHS information systems, the quality of lapsing data. To schedule a consult with an cyBoard@mail.mil) ding to the data consult |
| 10.6 Indicate how you will request data from | n the MHS. Select all that apply. |
| <ul> <li>□ Talking with MHS health care providers or MHS participants</li> <li>□ Obtaining MHS hard copy records specific to re</li> <li>☑ Obtaining data from an MHS information systematics</li> </ul> | esearch participants |
| | information system(s), indicate whether you p<br>cess an MHS information system directly to crea |
| A data extract is when the MHS or a contractor presearcher. When receiving a data set through dwhether the data elements should be provided as data extract, access to an information system med MHS information system and create a data set for Data Extract Access | ata extract, the researcher may indicate<br>s is, encrypted or collapsed. In contrast to a<br>eans that the researcher may directly access an |
| 10.8 Do you intend to request de-identified | data from the MHS in your research study? |
| There are different two methods for de-identifying 1) Safe Harbor Method: Removing all of the ident researcher does not have actual knowledge that t combination with other information to identify the 2) Statistical Method: An expert, with appropriate accepted statistical and scientific principles and m individually identifiable, determines that the data C Yes No | tifiers listed in Table 1 below, provided that the the remaining data can be used alone or in a individual who is the subject of the information a knowledge of and experience with generally nethods for rendering information not |
| 10.9 Indicate the MHS information system(s | s) from which you will seek to obtain data |
| If you do not know which system(s) contains the DoD Researchers on Using MHS Data or request of PrivacyBoard@mail.mil. Below is a list of commonly used MHS systems. It data is not listed below, list the name of the system: PHI Systems: | guidance from an MHS data expert at: <b>DHA.</b> f the system from which you seek to obtain |
| MHS Information System | Requesting Data |
| : AHLTA | : Yes |
| : CHCS | : No |

| PII-Only Systems: | | | |
|---|---|---|---|
| MHS Information Syste | em | Requesting Data | |
| No records have been a | added | | |
| De-Identified Data & 0 | Other Systems: | | |
| Information System | | Requesting Data | |
| No records have been a | added | | |
| 10.10 Do you intend to<br>outside of the M | o merge or otherwise of the Delay including other Delay | | |
| <ul><li>○ Yes, will merge data</li><li>⊙ No, will not merge da</li></ul> | ta | | |
| members of the<br>information sys<br>If you will merg | research participants<br>tems.<br>Je data, also indicate n<br>oyers, or household mo | that you will request<br>on-MHS data element | elatives, employers, or<br>from MHS hard copies o<br>s about research partic<br>n participants that you |
| Data Element(s) | MHS | Non-MHS Systems | MHS Hard Copies |
| 1. Names | | V | |
| 2. Postal address<br>with only town,<br>city, state and zip<br>code | | | |
| 3. Postal address with all geographic subdivisions smaller than a state, including street address, city, county, precinct, zip code and their equivalent geocodes, except for the initial three digits of a zip code if, according to the current publicly available data from the Bureau of Census: 1) the geographic unit formed by combining all zip codes with the same three initial digits contains more than 20,000 people; and 2) the initial three digits of a zip code for all such geographic | | | |

| l | 1 | 1 | 1 1 |
|---|---|---|---|
| units containing<br>20,000 or fewer<br>people is changed<br>to 000 | | | |
| 4. Dates including all elements (except year) directly related to an individual, including birth date, admission date, discharge date, and date of death | V | | |
| 5. Ages over 89 and all elements of dates (including year) indicative of such age, unless you will only request a single category of "age 90 or older" | | | |
| 6. Telephone<br>numbers | V | | |
| 7. Fax numbers | | | |
| 8. Electronic mail addresses | V | | |
| 9. Social Security<br>numbers (SSNs) | | | |
| 10. Medical record<br>numbers | | | |
| 11. Health plan<br>beneficiary numbers | | | |
| 12. Account numbers | | | |
| 13. Certificate<br>/license numbers | | | |
| 14. Vehicle identifiers and serial numbers, including license plate numbers | | | |
| | - | | |

| 15. Device identifiers and serial numbers | | | | |
|---|---|---|---|---|
| 16. Web Universal<br>Resource Locators<br>(URLs) | | | | |
| 17. Internet<br>Protocol (IP)<br>address numbers | | | | |
| 18. Biometric identifiers, including finger and voice prints | | | | |
| 19. Full-face<br>photographic<br>images and any<br>comparable images | | | | |
| 20. Any other unique identifying number, characteristic, or code (Diagnosis, DEERS ID, EDI-PI, Rank) | | <b>&gt;</b> | | |
| If you are obtaining SSN<br>be used | If you are obtaining SSNs, provide a justification as to why and explain why a substitute cannot be used | | | |
| 10.12 Do you believe small cell size, o | it is possible for the M<br>or any unique data ele | | entifiable because of tr | iangulation, a |
| Triangulation means using different data elements that are not themselves identifiable but that when combined can be used to identify an individual. For example, triangulation would use rank and race together to determine the identity of an individual with a particular health condition. Small cell size means that there is only a small number of eligible individuals that satisfy the category description. Guidance for acceptable cell size is available from the Centers for Medicare and Medicaid Services. For example, the rank category of four star generals with a particular diagnosis may be less than 30, so the rank category may need to be expanded to include lower ranks. | | | | |
| A unique data element includes any unique features that are not explicitly enumerated in the categories of data in rows 1 – 20 of the table above (in Section 10.10), but that could be used to identify an individual. Unique data elements include characteristics that are not themselves identifying, such as the rank of general or admiral, or a race or gender, but within the context of other information could be identifiable. | | | | |
| O Yes, I believe there is a reasonable possibility the MHS data will become identifiable No, I believe there is no reasonable possibility the MHS data will become identifiable | | | | |

| C Yes C No C N/A 10.14 Managing Data (Data Management and/or Sharing Plan) and/or Human Biological Specimens for this Study: Include in this section the plan for acquiring data (both electronic and hard copy), access during the study, data/specimen storage and length of time stored, shipment/transmission, and the plan for storage and final disposition at the conclusion of the study. Describe any data agreements in place for accessing data within and/or outside of your institution (e.g., Data Sharing Agreement, Data Use Agreement, Business Agreements, etc.) Acquiring Data The majority of participant data will be accrued via self-report questionnaire. We plan to retrieve diagnostic codes from their PT SOAP notes on AHLTA, and we will estruct and de-identify whole SOAP notes from a subgroup of randomly selected participants. We will also use CHCS and AHLTA to determine when a participant has or will receive their fourth PT session, but this is marely for scheduling follow-up, and will not be retained as data. Data Entry and Integrity: For data entered by participants into the REDCap surveys, we presume that participants responded correctly. All data collection tools completed on paper will be scanned and initially entered disk, occerate any inconsiderations research team members, who will mark the instrument as "Unvertified" in REDCap. The scanned forms will be transmitted to CAPT Grego Ziemike va SAPE, who will use them to verify the entered data, correct any inconsistencies, and them members, who will mark the instrument as "Complete". Our Excul database has been designed to draw values directly from downloaded REDCap data reports, rectuming the picture like for teams are mark We have access to the original data; de-identified data and endicientified SAP notes (for training evaluation) will be securely transmitted to them using the SAPE computer app. Data Storage. All physical data and consent forms will be maintained in locked cabinets within a locked office at MMCP, forms collected at branch clinics may | | |
|---|---|---|
| Include in this section the plan for acquiring data (both electronic and hard copy), access during the study, data/spectimen storage and length of time stored, shipment/transmission, and the plan for storage and final disposition at the conclusion of the study. Describe any data agreements in place for accessing data within and/or outside of your institution (e.g., Data Sharing Agreement, Data Use Agreement, Business Agreements, etc.) Acquiring Data. The majority of participent data will be accrued via self-report questionnaire. We plan to retrieve diagnostic codes from their PT SOAP notes on AHLTA, and we will extract and de-identify whole SOAP notes from a subgroup of randomly selected participants. We will also use CHCS and AHLTA to determine when a participant has or will receive their forth PT session, but this is most property for scheduling follow-up, and will not be retained as data. Data Entry and Integrity. For data entered by participants into the REDCap surveys, we presume that participants responded correctly. All data collection tools completed on paper will be scanned and initially entered and SECDcap by the procintoring research team member, who will mark the instrument as "Unvertified" in REDCap. The scanned forms will be transmitted to CAPT Gregg Ziemike via SAFE, who will use them to verify the entered data, correct any nonestistencies, and then mark the instrument as "Compiled." Our Excel database has been designed to draw values directly from downloaded REDCap data reports, reducing the potential for human error. We have also employed Excels conditional logic programming and formatting to alert us if a participant's records are incomplete or mismatched. Access to Data: The PI and research contractors (Gregg Ziemko and Timothy Hope) will have access to all study data, electronic and hard copy. NYII collaborators (Tr. Marco Campello and Dr. Sherri Wesser) will not have access to the original data; electionic and hard copy. NYII collaborators or the process of the stransmitted to them usin | O No | |
| the study, data/specimen storage and flend though the conclusion of the study. Describe any data as agreements in place for accessing data within and/or outside of your institution (e.g., Data Sharing Agreement, Data Use Agreement, Business Agreements, etc.) Acquiring Data: The majority of participant data will be accrued via self-report questionnaire. We plan to retrieve diagnostic codes from their PT SOAP notes on AHLTA, and we will extract and de-identify whole SOAP notes from a subgroup of randomly selected participants. We will also use CHCS and AHLTA to determine when a participant has or will receive their fourth PT session, but this is merely for scheduling follow-up, and will not be retained as data. Data Entry and Integrity. For data entered by participants into the REDCap surveys, we presume that participants responded correctly. All data collection tools completed on paper will be scanned and initially entered into REDCap by the proctoring research team member, who will mark the instrument as "Unvertified" in REDCap. The scanned forms will be transmitted to CAPT Grogg Ziemko via SAFE, who will use them to verify the entered data, correct any inconsistencies, and then mark the instrument as "Complete." Our Excel database has been designed to draw values directly from downloaded REDCap data reports, reducing the potential for human error. We have also employed Excel's conditional logic programming and formatting to alert us if a participant's records are incomplete or mismatched. Access to Data. The P1 and research contractors (Gregg Ziemke and Timothy Hope) will have access to all study data, electronic and hard copy. NYU collaborators (Dr. Marco Campello and Dr. Sherri Weiser) will not have access to the original data; de-identified data and de-identified SOAP notes (for training evaluation) will be securely transmitted to them NUC price. All digital data will be maintained in locked cabinets within a locked office at NMCP; forms collected at branch clinics may be temporarily stored in a smiler | | pecimens for |
| retrieve diagnostic codes from their PT SOAP notes on AHLTA, and we will extract and de-identify whole SOAP notes from a subgroup of randomly selected participants. We will also use CHCS and AHLTA to determine when a participant has or will receive their fourth PT session, but this is merely for scheduling follow-up, and will not be retained as data. Data Entry and Integrity: For data entered by participants into the REDCap surveys, we presume that participants responded correctly. All data collection tools completed on paper will be scanned and initially entered into REDCap by the proctoring research team member, who will mark the instrument as "Unverified" in REDCap. The scanned forms will be transmitted to CAPT Gregg Ziemke via SAFE, who will use them to verify the entered data, correct any inconsistencies, and them mark the instrument as "Complete." Our Excel database has been designed to draw values directly from downloaded REDCap data reports, reducing the potential for human error. We have also employed Excel's conditional logic programming and formatting to allert us if a participant's records are incomplete or mismatched. Access to Data: The PI and research contractors (Gregg Ziemke and Timothy Hope) will have access to all study data, electronic and hard copy, NYU collaborators (Dr. Marco Campello and Dr. Sherri Weiser) will not have access to the original data, de-identified data and de-identified SOAP notes (for training evaluation) will be securely transmitted to them using the SAFE computer app. Data Storage: All physical data and consent forms will be maintained in locked cabinets within a locked office at NMCP; froms collected at branch clinics may be temporarily stored in a similar two-lock situation until they can be transferred to the NMCP office, All digital data will be originally generated or collected on GFE at NMCP and maintained on that network. De-identified digital data will be originally generated or collected on GFE at NMCP and maintained on that network. De-identified digital d | the study, data/specimen storage and length of time stored, shipment/transmission, and the plan for storage and final disposition at the conclusion of the study. Describe any data agreements in place for accessing data within and/or outside of your institution (e.g., Data | |
| participants responded correctly. All data collection tools completed on paper will be scanned and initially entered into REDCap by the proctoring research team member, who will mark the instrument as "Unverified" in REDCap. The scanned forms will be transmitted to CAPT Gregg Ziemke via SAFE, who will use them to verify the entered data, correct any inconsistencies, and then mark the instrument as "Complete." Our Excel database has been designed to draw values directly from downloaded REDCap data reports, reducing the potential for human error. We have also employed Excel's conditional logic programming and formatting to alert us if a participant's records are incomplete or mismatched. Access to Data: The PI and research contractors (Gregg Ziemke and Timothy Hope) will have access to all study data, electronic and hard copy. NYU collaborators (Dr. Marco Campello and Dr. Sherri Weisser) will not have access to the original data; de-identified data and de-identified SOAP notes (for training evaluation) will be securely transmitted to them using the SAFE computer app. Data Storage: All physical data and consent forms will be maintained in locked cabinets within a locked office at NMCP; forms collected at branch clinics may be temporarily stored in a similar two-lock situation until they can be transferred to the NMCP office. All digital data will be originally generated or collected on GFE at NMCP and maintained on that network. De-identified digital data will be transmitted to the NYU collaborators. Shipment/Transmission: Any physical data that needs to be transferred from branch clinics to the NMCP office will be transported by a member of the NMCP research personnel. Transmission of digital data to NYU collaborators will be through the SAFE program. Conclusion: The investigators will maintain the de-identified data in a secure location for a period of six years after the end of the contract period. At the end of six years the de-identified subject questionnaire data will be destroyed. The PI will notify CD | retrieve diagnostic codes from their PT SOAP notes on AHLTA, and we will extract and de-identify whole SOAP notes from a subgroup of randomly selected participants. We will also use CHCS and AHLTA to determine when a participant has or will receive their fourth PT session, but this is merely for scheduling follow-up, and | |
| study data, electronic and hard copy. NYU collaborators (Dr. Marco Campello and Dr. Sherri Weiser) will not have access to the original data; de-identified data and de-identified SOAP notes (for training evaluation) will be securely transmitted to them using the SAFE computer app. Data Storage: All physical data and consent forms will be maintained in locked cabinets within a locked office at NMCP; forms collected at branch clinics may be temporarily stored in a similar two-lock situation until they can be transferred to the NMCP office. All digital data will be originally generated or collected on GFE at NMCP and maintained on that network. De-identified digital data will be transmitted to the NYU collaborators. Shipment/Transmission: Any physical data that needs to be transferred from branch clinics to the NMCP office will be transported by a member of the NMCP research personnel. Transmission of digital data to NYU collaborators will be through the SAFE program. Conclusion: The investigators will end support of dissemination of research data at the end of the project's contract period. The investigators will maintain the de-identified data in a secure location for a period of six years after the end of the contract period. At the end of six years the de-identified subject questionnaire data will be destroyed. The PI will notify CDMRP, the NMCP regulatory facilities such as IRB of record of the fulfillment of the requirement to destroy the research data at the end of the four and a half year period. Data Agreements: Once the protocol is approved, NYU will apply for a DHA Data Sharing Agreement, with NYU listed as the applicant/primary contractor and HJF staff listed as subcontractors. | participants responded correctly. All data collection tools completed on paper will be scanned and initially entered into REDCap by the proctoring research team member, who will mark the instrument as "Unverified" in REDCap. The scanned forms will be transmitted to CAPT Gregg Ziemke via SAFE, who will use them to verify the entered data, correct any inconsistencies, and then mark the instrument as "Complete." Our Excel database has been designed to draw values directly from downloaded REDCap data reports, reducing the potential for human error. We have also employed Excel's conditional logic programming and | |
| NMCP; forms collected at branch clinics may be temporarily stored in a similar two-lock situation until they can be transferred to the NMCP office. All digital data will be originally generated or collected on GFE at NMCP and maintained on that network. De-identified digital data will be transmitted to the NYU collaborators. Shipment/Transmission: Any physical data that needs to be transferred from branch clinics to the NMCP office will be transported by a member of the NMCP research personnel. Transmission of digital data to NYU collaborators will be through the SAFE program. Conclusion: The investigators will end support of dissemination of research data at the end of the project's contract period. The investigators will maintain the de-identified data in a secure location for a period of six years after the end of the contract period. At the end of six years the de-identified subject questionnaire data will be destroyed. The PI will notify CDMRP, the NMCP regulatory facilities such as IRB of record of the fulfillment of the requirement to destroy the research data at the end of the four and a half year period. Data Agreements: Once the protocol is approved, NYU will apply for a DHA Data Sharing Agreement, with NYU listed as the applicant/primary contractor and HJF staff listed as subcontractors. | study data, electronic and hard copy. NYU collaborators (Dr. Marco Campello and Dr. Sherri Weiser) will not have access to the original data; de-identified data and de-identified SOAP notes (for training evaluation) will be | |
| will be transported by a member of the NMCP research personnel. Transmission of digital data to NYU collaborators will be through the SAFE program. Conclusion: The investigators will end support of dissemination of research data at the end of the project's contract period. The investigators will maintain the de-identified data in a secure location for a period of six years after the end of the contract period. At the end of six years the de-identified subject questionnaire data will be destroyed. The PI will notify CDMRP, the NMCP regulatory facilities such as IRB of record of the fulfillment of the requirement to destroy the research data at the end of the four and a half year period. Data Agreements: Once the protocol is approved, NYU will apply for a DHA Data Sharing Agreement, with NYU listed as the applicant/primary contractor and HJF staff listed as subcontractors. | NMCP; forms collected at branch clinics may be temporarily stored in a similar two-lock situation until they can be transferred to the NMCP office. All digital data will be originally generated or collected on GFE at NMCP and | |
| contract period. The investigators will maintain the de-identified data in a secure location for a period of six years after the end of the contract period. At the end of six years the de-identified subject questionnaire data will be destroyed. The PI will notify CDMRP, the NMCP regulatory facilities such as IRB of record of the fulfillment of the requirement to destroy the research data at the end of the four and a half year period. Data Agreements: Once the protocol is approved, NYU will apply for a DHA Data Sharing Agreement, with NYU listed as the applicant/primary contractor and HJF staff listed as subcontractors. | will be transported by a member of the NMCP research personnel. Transmission of digital data to NYU | |
| listed as the applicant/primary contractor and HJF staff listed as subcontractors. | contract period. The investigators will maintain the de-identified data in a secure location for a period of six years after the end of the contract period. At the end of six years the de-identified subject questionnaire data will be destroyed. The PI will notify CDMRP, the NMCP regulatory facilities such as IRB of record of the | |

If the study involves collecting, storing, or banking human specimens, data, or documents (either by the Investigator or through an established repository) for FUTURE research, address.

Future Research:

How the specimens/data will be used, where and how data/specimens will be stored (including shipping procedures, storage plan, etc.), whether and how consent will be obtained, procedures that will fulfill subjects' request as stated in the consent, whether subjects may withdraw their data/specimens from storage, whether and how subjects may be recontacted for future research and given the option to decline, whether there will be genetic testing on the specimens, who will have access to the data/specimens, and the linkage, the length of time that data/specimens will be stored and conditions under which data/specimens will be destroyed.

N/A

# 11.0 Statistical/Data Analysis Plan

# 11.1 Statistical Considerations:

List the statistical methods to be used to address the primary and secondary objectives, specific aims, and/or research hypotheses. Explain how missing data and outliers will be handled in the analysis. The analysis plan should be consistent with the study objectives. Include any subgroup analyses (e.g., gender or age group). Specify statistical methods and variables for each analysis. Describe how confounding variables will be controlled in the data analysis

The characteristics of subjects including demographics and questionnaire responses will be summarized using descriptive statistics (e.g. mean ± standard deviation for continuous variables, and counts (%) for categorical variables). Alternatively, response frequencies for the questionnaires will be determined and displayed in tabular and graphic formats. After examining the response frequencies, some variable categories will be collapsed in order to allow further analysis using them as dependent measures in subsequent analysis (chi-square and logistic regression analyses). For the continuous outcomes (quantitative measurements such as Pain Disability Index scale, self-efficacy, positive outcome expectations, catastrophizing, fear avoidance beliefs and distress in Aims 2 and 3), we will conduct the Kolmogorov-Smirnov or the Shapiro-Wilk test to confirm the normality prior to performing statistical analyses. We will detect outliers via histograms, box-plots, normal plots and summary statistics. Where appropriate, we will conduct logarithmic transformation on variables.

All analyses will be conducted using the principle of "intent-to-treat" in which every participant is assumed to have received his/her assigned intervention, regardless of adherence.

# 11.2 Sample Size:

600

## 11.3 Total number of subjects requested (including records and specimens):

600

# 11.4 If you are recruiting by study arm, please identify the arms of the study and how many subjects will be enrolled in each arm

300 in the pre-training arm (control arm) 300 in the post-training arm (intervention arm)

# 11.5 Please provide a justification for your sample size

In order to achieve a statistical power of greater than 80% at an effect size of 0.3, we require a minimum of 200 participants to complete all follow-up in each cohort of the study, as detailed in the power analysis in Section 11.6. In order to account for a roughly 30% rate of attrition, we are requesting a sample size of 300 participants per arm, for a total of 600. Based on previous longitudinal studies by team members Dr. Campello, Dr. Weiser, and CAPT Ziemke, <sup>11,19,56,57</sup> we believe that this is a conservative estimate considering the duration of each participant's involvement.

# 11.6 Data Analysis Plan: Complete description: Background, Objectives, Design, Step by Step how the project is going to be done, Data analysis plan:

In order to assess for significant differences between two cohorts of patients, bivariate comparisons will first be conducted using a Chi-squared (Fisher exact) test to compare proportions of categorical (dichotomous outcomes) and an unpaired t-test for mean changes of continuous outcomes (i.e. Pain Disability Index scale, self-efficacy, positive outcome expectation, catastrophizing, fear avoidance beliefs and distress).

Alternatively, Wilcoxon nonparametric counterpart will be used for continuous variables where there is deviation from normality. These univariate analyses will be followed by multivariable regression methods for an adjustment of all other potential confounding variables. We will also use longitudinal logistic models (i.e., mixed-effects regression models with a random subject effect and GEE with exchangeable and independent correlations) to analyze the changes of the outcome at baseline at all follow-up times (baseline, post-treatment, at 6 months, and 1 year). Psychological outcomes will be analyzed at baseline and at post-treatment (approximately 4 weeks of enrollment). The models will be specified with random intercepts and slopes such that a linear trajectory representing outcomes will be compared between two arms. For example, longitudinal changes in all available continuous psychological outcomes over time of follow-up will be displayed using locally weighted smoothing scatter (lowess) plots, identifying nonparametric mean trajectories over time.<sup>86</sup> Mean trajectories then will be modeled with mixedeffects linear regression models, and if necessary using segment-linear models to approximate non-linear mean trajectories for ease of interpretation. Group (arm)-specific (as well as individual-level) intercepts and slopes over the period of follow-up will be included as random effects, while other covariates such as other clinical or demographic confounders will be modeled as fixed effects. An interaction term will be also assessed to test group differences in outcomes over time. Residual-based diagnostics will be used to evaluate validity of model assumptions. Two sided p-values <0.05 will be considered to be statistically significant. All statistical procedures will be performed using R statistical package (www.R-project.org).

In order to determine the association of treatment effects among the subjects who endorse the mental care questions, we will further perform the sub-analysis using the regression analysis similarly stated as above. All covariates and their source are shown in the tables of variables found in Section 10.2. This analytic approach will be hypotheses generating and will be largely exploratory as the study may not be powered to detect significant effects. Therefore, we have not proposed any formal power calculation for the sub-analysis.

Assuming normality, we calculated the statistical power for various detectable effect sizes and sample sizes in a two-sided hypothesis test with a significance level of 0.05, where the ratio of sample size of 1:1 is assumed between cases (intervention arm) vs. controls. When outcomes are proportions, we calculated power based on rate differences. Table 2 shows that our sample size will have adequate power to detect listed effect sizes. For example, we will achieve 95.4% power to detect a difference of rate of 0.3 (i.e., achieving minimal clinically important difference of 80% in receiving therapy by PT staff "after training" group vs. 50% in receiving therapy by PT staff before training) between two arms of a size of 100 (117) for each with 30 (40) % of missingness. For continuous outcomes, the same size of n=100 (117) for each will have a 83.6% power to detect standardized mean difference of 0.5, which corresponds that the reduction in PDI (Pain Disability Index) score from baseline to follow-up would be 50% greater in the training group as compared to that before training. Note that for each domain outcome, the power is the same for each effect size since they are standardized, but the mean change corresponding to a given effect size differs.

| Table 2. Sa | Table 2. Sample size and power | | | | |
|---|---|---|---|---|---|
| Cohort size<br>N<br>(Total<br>sample) | Loss to follow-up or<br>noncompliance | Unpaired t-<br>test | | Fisher exact test | |
| | | Effect size <sup>1</sup> | Power<br>(%) | Effect size <sup>2</sup> | Power<br>(%) |
| 117 (234)<br>100 (200) | 40%<br>30% | 0.5 | 83.6 | 0.30<br>(p1=0.8, p2=0.50) | 95.4 |
| 167 (334)<br>143 (286) | 40%<br>30% | 0.5 | 94 | 0.25<br>(p1=0.8, p2=0.55) | 95.8 |
| 250 (500)<br>215 (430) | 40%<br>30% | 0.4 | 93.2 | 0.20<br>(p1=0.8, p2=0.6) | 96 |
| 334 (668)<br>286 (572) | 40%<br>30% | 0.3 | 84.9 | 0.15<br>(p1=0.8, p2=0.<br>65) | 96 |

1 standardized mean difference of 2 groups
2 absolute proportion difference of 2 groups with proportions (p1=P(above MID in pre-training cohort), p2= p2=P(above MID in post-training cohort))

Missing data: We will make every effort to prevent and avoid missing data. Even with the most robust processes, however, some missing data is inevitable. We will assess the mechanism of missing data by comparing patients with and without missing values on baseline and other complete information, to detect any patterns in demographics or other characteristics associated with missing data. First, the various missingness assumptions (missing completely at random: MCAR, missing at random: MAR or missing not at random: MNAR) will be tested by comparing subjects with missing and non-missing data.87 In order to incorporate uncertainty in handling missing data, we will perform a multiple imputation, which begins with a prediction of the missing data using the existing data from other variables.88 The missing values will then be replaced with the predicted values, and a full data set called the imputed data set will be created. This process iterates the repeatability and makes multiple imputed data sets. Each multiple imputed data set produced will be then analyzed using the standard statistical analysis procedures for complete data, and give multiple analysis results. Subsequently, by combining these analysis results, a single overall analysis result will be produced.

| 12.0 Participant Information |
|---|
| 12.1 Subject Population: |
| US active duty service members receiving physical therapy for musculoskeletal disorders at Naval Medical Center Portsmouth and its branch health clinics. |
| 12.2 Age Range: |
| Check all the boxes that apply. if the age range of potential subjects (specimens, records) does not match the range(s) selected, please specify in the text box. 0-17 |
| ✓ Male ✓ Female ✓ Other |
| 12.4 Special categories, check all that apply |
| Minors /Children Students Employees - Civilian Employees - Contractor Resident/trainee Cadets /Midshipmen |
| Active Duty Military Personnel |
|---|
| ■ Wounded Warriors |
| Economically Disadvantaged Persons |
| Educationally Disadvantaged Persons |
| Physically Challenged (Physical challenges include visual and/or auditory impairment) |
| Persons with Impaired Decisional Capacity |
| Prisoners |
| ☐ Pregnant Women, Fetuses, and Neonates |
| □ Non-English Speakers |
| ☐ International Research involving Foreign Nationals - Headquarters Review is necessary |
| You must also consider the requirements of DoDI 3216.02, Enclosure 3, paragraph 7.e. |

# 12.5 Inclusion Criteria:

| Order<br>Number | Criteria |
|---|---|
| 1 | Active duty service members (at baseline; separation from the military post-treatment will not be grounds for exclusion) |
| 2 | Patients presenting to an NMCP or branch clinic physical therapy department |
| 3 | Patients who have only received their evaluation appointment for their primary complaint |
| 4 | Patients presenting for a primary complaint of a MSD (The following ICD-10 codes will be included: M13,M14.8,M15-19,M21-25,M40-43,M46-48,M50- 54,M60-71, M73,M75-77) |

# 12.6 Exclusion Criteria:

| Order<br>Number | Criteria |
|---|---|
| 1 | Patients not eligible to receive outpatient physical therapy. |
| 2 | Patients receiving fewer than four treatment sessions of physical therapy. |
| 3 | Patients who are pregnant |
| 4 | Patients receiving physical therapy for acute post-surgical recovery |
| 5 | Patients scheduled for or subject to a Physical Evaluation Board (PEB) at baseline |
| 6 | Coast Guard, as they are DoT rather than DoD |

# 13.0 Recruitment and Consent

13.1 Please describe the recruitment process, including how subjects will be identified and selected for the study.

| Research staff will approach pre-screened patients immediately after their evaluation appointment with their physical therapist, inform them of the study, and ask them if they are interested in participating. Interested patients will then be lead to a private study area nearby to begin the consenting process described in Section 13.4. Those who consent will leave us their contact information and may complete their baseline questionnaire immediately on location, or they may complete it remotely before their next appointment. | |
|---|---|
| 13.2 Compensation for Participation: | |
| Participants will not be compensated for participation. | |
| 13.3 Please describe the pre-screening process. If no pre-screening, enter Not Applicable i | n the text editor |
| Physical therapy staff will be informed of the inclusion and exclusion criteria for our study. Researchers will use printouts of the clinic schedule received from the clinic manager to determine which patients are coming in for evaluation. In Phase II, we will also use the schedule to verify that the patient's therapist has completed PiPT training. We will let staff members conducting evaluations know that we are interested in approaching their patients after the evaluation if they are eligible. If the staff member assents, we will brief the patient on the study and ask them to verify that they are: 1. An active duty service member beginning physical therapy for their current musculoskeletal injury 2. NOT pregnant, receiving PT for post-surgical follow-up, or scheduled for or subject to a Physical Evaluation Board. | |
| 13.4 Consent Process: Revised Common Rule, Section 219.116: General requirements for consent, whether written or oral, are set forth in this paragraph and apply to consent accordance with the requirements set forth in paragraphs (b) through (d) of this sect consent may be obtained in lieu of informed consent obtained in accordance with para (c) of this section only with respect to the storage, maintenance, and secondary reseat identifiable private information and identifiable biospecimens. | obtained in<br>ion. Broad<br>agraphs (b) and |
| Are you requesting a waiver or alteration of informed consent? | |
| O Yes ⊙ No | |
| tes to No | |
| Please explain the consent process: | |
| Please explain the consent process: Once patients have been prescreened and approached, patients will be shown to a private room to review the consent form with the researcher. The researcher will lead patients through the consent form using proper consenting procedures, then give patients time to further review the consent form privately and receive answers to any questions they may have regarding the study. Patients will be granted as much time as they need to make their decision in a private space. The patient will decide whether to participate, and will sign and date the consent form along with the researcher. The | |
| Please explain the consent process: Once patients have been prescreened and approached, patients will be shown to a private room to review the consent form with the researcher. The researcher will lead patients through the consent form using proper consenting procedures, then give patients time to further review the consent form privately and receive answers to any questions they may have regarding the study. Patients will be granted as much time as they need to make their decision in a private space. The patient will decide whether to participate, and will sign and date the consent form along with the researcher. The participant will also receive a duplicate copy of the consent form, signed and dated by the researcher. 13.5 DoDI 3216.02 requires an ombudsman to be present during recruitment briefings whe involves greater than minimal risk and recruitment of Service members occurs in a greater than minimal risk and recruitment of Servi | |
| Please explain the consent process: Once patients have been prescreened and approached, patients will be shown to a private room to review the consent form with the researcher. The researcher will lead patients through the consent form using proper consenting procedures, then give patients time to further review the consent form privately and receive answers to any questions they may have regarding the study. Patients will be granted as much time as they need to make their decision in a private space. The patient will decide whether to participate, and will sign and date the consent form along with the researcher. The participant will also receive a duplicate copy of the consent form, signed and dated by the researcher. 13.5 DoDI 3216.02 requires an ombudsman to be present during recruitment briefings who involves greater than minimal risk and recruitment of Service members occurs in a grapplicable, you may nominate an individual to serve as the ombudsman. | |

Explain the process for withdrawal and specify whether or not the subjects will be given the opportunity to withdraw their data their data/specimens in the event they wish to withdraw from the study

Participants may contact a member of the research team using any of the contact methods on the ICF to let them know that they wish to withdraw. They will be prompted to revoke their HIPAA Authorization as well, and have instructions recapitulated.

Once we have received the participant's revocation of HIPAA Authorization, their data will be purged from the study.

## 14.0

# **Risks and Benefits**

## 14.1

## **Risks of Harm:**

Identify all research-related risks of harm to which the subject will be exposed for each research procedure or intervention as a result of participation in this study. Consider the risks of breach of confidentiality, psychological, legal, social, and economic risks as well as physical risks. Do not describe risks from standard care procedures; only describe risks from procedures done for research purposes

As with most studies, there is a risk of breaches of privacy and/or confidentiality.

Additionally, during our initial questionnaire we ask our participants to self-report on a number of psychological and social health measures, notably depression, anxiety, and PTSD. It is possible that some participants may become distressed while answering these questions. If a participant experiences an emergent mental health event, the researcher will immediately contact a clinician to transfer the patient to the Emergency Medicine Department (EMD).

## 14.2

## Measures to Minimize Risks of Harm (Precautions, safeguards):

For each research procedure or intervention, describe all measures to minimize and/or eliminate risk of harms to subjects and study personnel

We will minimize risks of confidentiality and privacy breaches as described in Sections 14.3 and 14.5, respectively.

We will address the potential for distress by informing patients of the nature of the questionnaires during the consenting process. Additionally, the survey tools we use to measure aspects of mental health are established, validated clinical psychology measures. If a participant grows distressed while responding to the questionnaire, we will notify their physical therapist, who may refer them to the adult mental health department or the emergency department, depending on the severity and urgency of the incident.

## 14.3

# Confidentiality Protections (for research records, data and/or specimens):

Describe in detail the plan to maintain confidentiality of the research data, specimens, and records throughout the study and at its conclusion (e.g., destruction, long term storage, or banking). Explain the plan for securing the data (e.g., use of passwords, encryption, secure servers, firewalls, and other appropriate methods). If data will be shared electronically with other team members/collaborators outside the institution, describe the method of transmission and safeguards to maintain confidentiality. Explain whether this study may collect information

that State or Federal law requires to be reported to other officials or ethically requires action, e. q., child or spouse abuse

Electronic study data will primarily be housed on government furnished equipment, and files containing PII will be password protected. All data transmitted to NYU personnel will be deidentified and transmitted via SAFE. Paper forms such as consent forms and questionnaires will be secured in locked cabinets behind at least one additional locked door. The consent forms and intake forms, which contain identifiers, will be stored in a separate cabinet from any paper questionnaires.

We will be collecting data on distress, depression, anxiety, and PTSD. While any one of these measures may not be reportable, if our team psychologist believes these indicate a dangerous situation, e.g. a suicide risk, we will report to the appropriate authorities.

## 14.4

## **Potential Benefits:**

Describe any real and potential benefits of the research to the subject and any potential benefits to a specific community or society

If the individuals in the research are considered experimental subjects (per 10 USC 980), and they cannot provide their own consent, the protocol must describe the intent to directly benefit all subjects

Participants will not directly benefit, but we expect to improve physical therapy for ADSM with musculoskeletal disorders.

## 14.5

# **Privacy for Subjects:**

Describe the measures to protect subject's privacy during recruitment, the consent process, and all research activities, etc.

Recruiting and consenting: We intend to rely on physical therapy staff to introduce us to eligible patients in their exam room after their evaluation session, so that participants can be briefed on the study in private. Interested patients will be provided a private space in the PT clinic to review the consent form and ask questions.

Participation: Participants may either complete their baseline questionnaire in person or online; all follow-up questionnaires will be completed remotely. If they choose to participate in person, they will complete the questionnaire in paper in the consenting area. The online method will consist of the research team sending a link to the online questionnaire via encrypted email to the address specified by the participant. The online questionnaire will be hosted on REDCap.

## 14.6

## **Incidental or Unexpected Findings:**

Describe the plan to address incidental findings and unexpected findings about individuals from screening to the end of the subject's participation in the research. In cases where the subject could possibly benefit medically or otherwise from the information, state whether or not the results of screening, research participation, research tests, etc., will be shared with subjects or their primary care provider. State whether the researcher is obligated or mandated to report results to appropriate military or civilian authorities and explain the potential impact on the subject

While our study is observational and physical therapy is a lower-risk clinic, we will be viewing SOAP notes and administering mental health survey tools. Several members of our research team are physical therapists, and another is a psychologist. This puts us in a position to discover incidental findings of a two different natures.

Misdiagnosis or mistreatment of MSD: If the physical therapists on the research team conclude that a subject's MSD has been misdiagnosed or that their course of treatment is grossly inappropriate, they will pass that information along to the department head of physical therapy, so the matter can be brought to the attention of the participant's therapist. However, we only plan to do this if the patient is at risk of harm, not if the study team simply believes the course of treatment is sub-optimal.

Mental Health dangers: During our initial questionnaire, we ask our participants to self-report on a number of psychological and social health measures, notably PTSD, depression, and anxiety. If a participant scores >50 on the PCL-M scale for post-traumatic stress disorder, >16 on the CES-D scale for clinical depression, or >10 on the GAD-7 scale for anxiety disorder (the thresholds for severe psychiatric disorder) at baseline, we will notify the participant's physical therapist and our research monitor to make a referral for appropriate treatment. If we find evidence of an emergent mental health issue, a researcher will immediately contact the participant's physical therapist to transfer the patient to the Emergency Medicine Department (EMD).

# 15.0

# **Study Monitoring**

| 15.1 | Your study requires either Data and Safety Monitoring Plan (DSMP) or a Data and Safety Monitoring |
|---|---|
| | Board (DSMB). |

O DSMP

C DSMB

C Both

Not Applicable

# 16.0

## Reportable Events

16.1 Reportable Events: Consult with the research office at your institution to ensure requirements are met. Describe plans for reporting unexpected adverse events and unanticipated problems. Address how unexpected adverse events will be identified, who will report, how often adverse events and unanticipated problems will be reviewed to determine if any changes to the protocol or consent form are needed and the scale that will be used to grade the severity of the adverse event.

Consult with the research office at your institution to ensure requirements are met

- Describe plans for reporting expected adverse events. Identify what the expected adverse events will be for this study, describe the likelihood (frequency, severity, reversibility, short-term management and any long-term implications of each expected event)
- Describe plans for reporting unexpected adverse events and unanticipated problems. Address how unexpected adverse events will be identified, who will report, how often adverse events and unanticipated problems will be reviewed to determine if any changes to the research protocol or consent form are needed and the scale that will be used to grade the severity of the adverse event

We believe that the most likely adverse events are already described under "Incidental Findings" (Section 14.6). Beyond those, the most plausible adverse events we foresee are possible breaches of privacy and/or confidentiality and the potential distress of answering questions regarding mental health, which are also previously explored in Section 14.1.

reported within five business days. Other events such as non-serious adverse events and protocol deviations will be reported with the next continuing review unless they require a protocol modification. In that instance, the event will be reported alongside the modification. Research staff will inquire whether any adverse events (AEs) have occurred at each in-person encounter with participants, and REDCap surveys will include instructions for contacting the research coordinator or PI if an AE has occurred. All research staff interacting with participants will maintain blank AE Log forms. Due to the large sample size and low risk, an AE Log will not be maintained for every participant, only those involved in an AE. 17.0 **Equipment/non-FDA Regulated Devices** 17.1 Does the study involve the use of any unique non-medical devices/equipment? C Yes C No 18.0 **FDA-Regulated Products** 18.1 Will any drugs, dietary supplements, biologics, or devices be utilized in this study? □ Drugs Dietary Supplements ■ Biologics □ Devices ✓ N/A 18.5 Sponsor (organization/institution/company): ✓ N/A If applicable, provide sponsor contact information: 19.0 **Research Registration Requirements** 19.1 ClinicalTrials.gov Registration: Registration is not required Registration pending C Registration complete 19.2 Defense Technical Information Center Registration (Optional): Registration is not required Registration pending

C Registration complete

Any reportable events, expected or not, will result in our team submitting a Note to File to the IRB within 24 hours of discovery. Serious adverse events and unanticipated problems will be reported to the Research Subject Protection Division within 24 hours. Similarly, any protocol violations will be

#### 20.1 References:

- 1. Cohen, S. P., Nguyen, C., Kapoor, S. G., Anderson-Barnes, V. C., Foster, L., Shields, C., . . . Plunkett, A. (2009). Back pain during war: an analysis of factors affecting outcome. *Archives of internal medicine*, 169(20), 1916-1923.
- 2. Goodman, G. P., DeZee, K. J., Burks, R., Waterman, B. R., & Belmont, P. J. (2011). Epidemiology of psychiatric disorders sustained by a US Army brigade combat team during the Iraq War. *General hospital psychiatry*, 33(1), 51-57.
- 3. Huang, G. D. (2001). Back and upper extremity disorders among enlisted US Marines: burden and individual risk factors. *Military medicine*, 166(11), 1007.
- 4. Patzkowski, J. C., Rivera, J. C., Ficke, J. R., & Wenke, J. C. (2012). The changing face of disability in the US Army: the Operation Enduring Freedom and Operation Iraqi Freedom effect. *J ournal of the American Academy of Orthopaedic Surgeons*, 20, S23-S30.
- 5. Belmont, P. J., Owens, B. D., & Schoenfeld, A. J. (2016). Musculoskeletal injuries in Iraq and

Afghanistan: epidemiology and outcomes following a decade of war. *Journal of the American Academy of Orthopaedic Surgeons*, 24(6), 341-348.

- 6. Cohen, S. P., Brown, C., Kurihara, C., Plunkett, A., Nguyen, C., & Strassels, S. A. (2010). Diagnoses and factors associated with medical evacuation and return to duty for service members participating in Operation Iraqi Freedom or Operation Enduring Freedom: a prospective cohort study. *Lancet*. 375. doi:10.1016/s0140-6736(09)61797-9
- 7. Shaffer, R. A., Brodine, S. K., Ito, S. I., & Le, A. T. (1999). Epidemiology of illness and injury among US Navy and Marine Corps female training populations. *Military medicine*, 164(1), 17.
- 8. Bohnker, B. K., Telfair, T., McGinnis, J. A., Malakooti, M. A., & Sack, D. M. (2003). Analysis of Navy physical evaluation board diagnoses (1998-2000). *Military medicine*, 168(6), 482.
- 9. Hebert, D. J., & Pasque, C. B. (2004). Orthopedic injuries during carrier battle group deployments. *Mil Med*, 169(3), 176-180. doi:10.7205/milmed.169.3.176
- 10. Lewis Shattuck, N., Matsangas, P., Moore, J., & Wegemann, L. (2016). Prevalence of Musculoskeletal Symptoms, Excessive Daytime Sleepiness, and Fatigue in the Crewmembers of a U.S. Navy Ship. *Military medicine*, 181(7), 655-662. doi:10.7205/milmed-d-15-00279
- 11. Weiser, S., Lis, A., Brennan, T., Ziemke, G., Hievert, R., Iveson, B., . . . Campello, M. (2019). What do patients learn from psychologically based physical therapy? . *Journal of Physical Therapy Education*.
- 12. Ziemke, G., Campello, M., Hiebert, R., Weiner, S. S., Rennix, C., & Nordin, M. (2015). Does Coordinated, Multidisciplinary Treatment Limit Medical Disability and Attrition Related to Spine Conditions in the US Navy? *Clin Orthop Relat Res*, 473(9), 2920-2928. doi:10.1007/s11999-015-4328-4
- 13. Feuerstein, M., Berkowitz, S. M., & Peck Jr, C. A. (1997). Musculoskeletal-related disability in US Army personnel: prevalence, gender, and military occupational specialties. Journal of occupational and environmental medicine, 39(1), 68-78.
- 14. Berkowitz, S. M. (1999). Occupationa back disability in US Army personnel. *Military medicine*, 164(6), 412.
- 15. Lincoln, A. E., Smith, G. S., Amoroso, P. J., & Bell, N. S. (2002). The natural history and risk factors of musculoskeletal conditions resulting in disability among US Army personnel. *Work*, 18.
- 16. Schoenfeld, A. J., Goodman, G. P., Burks, R., Black, M. A., Nelson, J. H., & Belmont, P. J., Jr. (2014). The Influence of Musculoskeletal Conditions, Behavioral Health Diagnoses, and Demographic Factors on Injury-Related Outcome in a High-Demand Population. *J Bone Joint Surg Am*, 96(13), e106.

doi:10.2106/jbjs.M.01050

- 17. Booth-Kewley, S., Larson, G. E., & Highfill-McRoy, R. M. (2009). Psychosocial predictors of return to duty among marine recruits with musculoskeletal injuries. *Military Medicine*, 174(2), 139-152. doi:10.7205/milmed-d-01-2708
- 18. Booth-Kewley, S., Schmied, E. A., Highfill-McRoy, R. M., Sander, T. C., Blivin, S. J., & Garland, C. F. (2014). A prospective study of factors affecting recovery from musculoskeletal injuries. *J Occup Rehabil*, 24(2), 287-296. doi:10.1007/s10926-013-9456-7
- 19. Hiebert, R., Campello, M. A., Weiser, S., Ziemke, G. W., Fox, B. A., & Nordin, M. (2012). Predictors of short-term work-related disability among active duty US Navy personnel: a cohort study in patients with acute and subacute low back pain. The Spine Journal, 12(9), 806-816.
- 20. Hodges, P. W., & Richardson, C. A. (1996). Inefficient muscular stabilization of the lumbar spine associated with low back pain. A motor control evaluation of transversus abdominis. *Spine* (Phila Pa 1976), 21(22), 2640-2650. doi:10.1097/00007632-199611150-00014
- 21. Ferreira, P. H., Ferreira, M. L., Maher, C. G., Refshauge, K., Herbert, R. D., & Hodges, P. W. (2010). Changes in recruitment of transversus abdominis correlate with disability in people with chronic low back pain. *Br J Sports Med*, 44(16), 1166-1172. doi:10.1136/bjsm.2009.061515
- 22. Sudhaus, S., Mollenberg, T., Plaas, H., Willburger, R., Schmieder, K., & Hasenbring, M. (2012). Cortisol awakening response and pain-related fear-avoidance versus endurance in patients six months after lumbar disc surgery. *Appl Psychophysiol Biofeedback*, 37(2), 121-130. doi:10.1007/s10484-012-9186-1
- 23. Dawson, A. P., Schluter, P. J., Hodges, P. W., Stewart, S., & Turner, C. (2011). Fear of movement, passive coping, manual handling, and severe or radiating pain increase the likelihood of sick leave due to low back pain. *Pain*, 152(7), 1517-1524. doi:10.1016/j.pain.2011.02.041
- 24. Kendall, N A S,Linton, S J & Main, C J (1997). Guide to Assessing Psycho-social Yellow Flags in Acute Low Back Pain: RiskFactors for Long-Term Disability and Work Loss. Accident Compensation Corporation and the New ZealandGuidelines Group, Wellington, New Zealand. (Oct, 2004 Edition).
- 25. Nicholas, M. K., Linton, S. J., Watson, P. J., & Main, C. J. (2011). Early identification and management of psychological risk factors ("yellow flags") in patients with low back pain: a reappraisal. *Phys Ther*, 91(5), 737-753. doi:10.2522/ptj.20100224
- 26. Wertli, M. M., Held, U., Lis, A., Campello, M., & Weiser, S. (2018). Both positive and negative beliefs are important in patients with spine pain: findings from the Occupational and Industrial Orthopaedic Center registry. Spine J, 18(8), 1463-1474. doi:10.1016/j.spinee.2017.07.166
- 27. Keefe, F. J., Beaupre, P. M., Gil, K. M., Rumble, M. E., & Aspnes, A. K. (1996). Group therapy for patients with chronic pain. . *In Pain Management: A Practitioner's Handbook* (Vol. 2, pp. 234-255).
- 28. Turk, D. C., Meichenbaum, D., & Genest, M. (1987). *Pain and Behavioral Medicine: A Cognitive-Behavioral Perspective*. New York, NY: The Guilford Press.
- 29. Foster, N. E., & Delitto, A. (2011). Embedding psychosocial perspectives within clinical management of low back pain: integration of psychosocially informed management principles into physical therapist practice--challenges and opportunities. *Phys Ther*, 91(5), 790-803. doi: 10.2522/ptj.20100326
- 30. Main, C. J., Foster, N., & Buchbinder, R. (2010). How important are back pain beliefs and expectations for satisfactory recovery from back pain? *Best Pract Res Clin Rheumatol*, 24(2), 205-217.
- doi:10.1016/j.berh.2009.12.012
- 31. Hoffman, S. G. (2011). An Introduction to Modern CBT: Psychological Solutions to MEntal Health Problems: John Wiley & Sons.
- 32. Nicholas, M. K., & George, S. Z. (2011). Psychologically informed interventions for low back pain: an update for physical therapists. *Phys Ther*, 91(5), 765-776. doi:10.2522/ptj.20100278
- 33. Shaw, W. S., van der Windt, D. A., Main, C. J., Loisel, P., & Linton, S. J. (2009). Early patient screening and intervention to address individual-level occupational factors ("blue flags") in back disability. *J Occup Rehabil*, 19(1), 64-80. doi:10.1007/s10926-008-9159-7
- 34. Wertli, M. M., Rasmussen-Barr, E., Weiser, S., Bachmann, L. M., & Brunner, F. (2014). The role of fear avoidance beliefs as a prognostic factor for outcome in patients with nonspecific low back pain: a systematic review. *Spine J*, 14(5), 816-836.e814. doi:10.1016/j.spinee.2013.09.036

- 35. Foster, N. E., Mullis, R., Young, J., Doyle, C., Lewis, M., Whitehurst, D., & Hay, E. M. (2010). IMPaCT Back study protocol. Implementation of subgrouping for targeted treatment systems for low back pain patients in primary care: a prospective population-based sequential comparison. *B MC Musculoskelet Disord*, 11, 186. doi:10.1186/1471-2474-11-186
- 36. Vlaeyen, J. W. S., Maher, C. G., Wiech, K., Van Zundert, J., Meloto, C. B., Diatchenko, L., . . Linton, S. J. (2018). Low back pain. *Nat Rev Dis Primers*, 4(1), 52. doi:10.1038/s41572-018-0052-1
- 37. Karjalainen, K., Malmivaara, A., Pohjolainen, T., Hurri, H., Mutanen, P., Rissanen, P., . . . Roine, R. (2003). Mini-intervention for subacute low back pain: a randomized controlled trial. *Spi* ne, 28(6), 533-540.
- 38. Hayden, J. A., van Tulder, M. W., Malmivaara, A. V., & Koes, B. W. (2005). Meta-analysis: exercise therapy for nonspecific low back pain. Ann Intern Med, 142(9), 765-775.
- 39. Keller, A., Hayden, J., Bombardier, C., & Van Tulder, M. (2007). Effect sizes of non-surgical treatments of non-specific low-back pain. *European Spine Journal*, 16(11), 1776-1788.
- 40. Herman, P. M., Anderson, M. L., Sherman, K. J., Balderson, B. H., Turner, J. A., & Cherkin, D. C. (2017). Cost-effectiveness of Mindfulness-based Stress Reduction Versus Cognitive Behavioral Therapy or Usual Care Among Adults With Chronic Low Back Pain. *Spine* (Phila Pa 1976), 42(20), 1511-1520. doi:10.1097/brs.0000000000002344
- 41. Chou, R., Deyo, R., Friedly, J., Skelly, A., Hashimoto, R., Weimer, M., . . . Brodt, E. D. (2017).

Nonpharmacologic Therapies for Low Back Pain: A Systematic Review for an American College of Physicians Clinical Practice Guideline. *Ann Intern Med*, 166(7), 493-505. doi:10.7326/m16-2459

- 42. Lamb, S. E., Hansen, Z., Lall, R., Castelnuovo, E., Withers, E. J., Nichols, V., . . . investigators, B. S. T. T. (2010). Group cognitive behavioural treatment for low-back pain in primary care: a randomized controlled trial and cost-effectiveness analysis. *The Lancet*, 375 (9718), 916-923.
- 43. Burton, A. K., Balague, F., Cardon, G., Eriksen, H. R., Henrotin, Y., Lahad, A., . . . van der Beek, A. J. (2006). Chapter 2. European guidelines for prevention in low back pain: November 2004. *Eur Spine J*, 15 Suppl 2, S136-168. doi:10.1007/s00586-006-1070-3
- 44. van der Windt, D., Hay, E., Jellema, P., & Main, C. (2008). Psychosocial interventions for low back pain in primary care: lessons learned from recent trials. *Spine* (Phila Pa 1976), 33(1), 81-89.

## doi:10.1097/BRS.0b013e31815e39f9

- 45. Main, C. J., & George, S. Z. (2011). Psychologically informed practice for management of low back pain: future directions in practice and research. *Phys Ther*, 91(5), 820-824. doi:10.2522/ptj. 20110060
- 46. Sanders, T., Foster, N. E., Bishop, A., & Ong, B. N. (2013). Biopsychosocial care and the physiotherapy encounter: physiotherapists' accounts of back pain consultations. *BMC musculoskeletal disorders*, 14(1), 65. doi:10.1186/1471-2474-14-65
- 47. Synnott, A., O'Keeffe, M., Bunzli, S., Dankaerts, W., O'Sullivan, P., & O'Sullivan, K. (2015).

Physiotherapists may stigmatise or feel unprepared to treat people with low back pain and psychosocial factors that influence recovery: a systematic review. *J Physiother*, 61(2), 68-76.

## doi:10.1016/j.jphys.2015.02.016

- 48. Bryant, C., Lewis, P., Bennell, K. L., Ahamed, Y., Crough, D., Jull, G. A., . . . Keefe, F. J. (2014). Can physical therapists deliver a pain coping skills program? An examination of training processes and outcomes. *Physical Therapy*, 94(10), 1443-1454.
- 49. Nielsen, M., Keefe, F. J., Bennell, K., & Jull, G. A. (2014). Physical therapist-delivered cognitivebehavioral therapy: a qualitative study of physical therapists' perceptions and experiences. *Phys Ther*, 94(2), 197-209. doi:10.2522/ptj.20130047
- 50. Jacobs, C. M., Guildford, B. J., Travers, W., Davies, M., & McCracken, L. M. (2016). Brief

psychologically informed physiotherapy training is associated with changes in physiotherapists' attitudes and beliefs towards working with people with chronic pain. *Br J Pain*, 10(1), 38-45.

# doi:10.1177/2049463715600460

- 51. Beneciuk, J. M., George, S. Z., Greco, C. M., Schneider, M. J., Wegener, S. T., Saper, R. B., & Delitto, A. (2019). Targeted interventions to prevent transitioning from acute to chronic low back pain in highrisk patients: development and delivery of a pragmatic training course of psychologically informed physical therapy for the TARGET trial. *Trials*, 20(1), 256. doi:10.1186/s13063-019-3350-3
- 52. Hunt, M. A., Keefe, F. J., Bryant, C., Metcalf, B. R., Ahamed, Y., Nicholas, M. K., & Bennell, K. L. (2013). A physiotherapist-delivered, combined exercise and pain coping skills training intervention for individuals with knee osteoarthritis: a pilot study. *Knee*, 20(2), 106-112. doi: 10.1016/j.knee.2012.07.008
- 53. Pincus, T., Anwar, S., McCracken, L. M., McGregor, A., Graham, L., Collinson, M., . . . Farrin, A. J. (2015). Delivering an Optimised Behavioural Intervention (OBI) to people with low back pain with high psychological risk; results and lessons learnt from a feasibility randomised controlled trial of Contextual Cognitive Behavioural Therapy (CCBT) vs. Physiotherapy. *BMC Musculoskelet Disord*, 16, 147.

# doi:10.1186/s12891-015-0594-2

- 54. Archer, K. R., Coronado, R. A., & Wegener, S. T. (2018). The Role of Psychologically Informed Physical Therapy for Musculoskeletal Pain. *Current Physical Medicine and Rehabilitation Reports*, 6(1), 15-25.
- 55. Overmeer, T., Boersma, K., Denison, E., & Linton, S. J. (2011). Does Teaching Physical Therapists to Deliver a Biopsychosocial Treatment Program Result in Better Patient Outcomes? A Randomized Controlled Trial. Physical Therapy, 91(5), 804-819. doi:10.2522/ptj.20100079
- 56. Campello, M., Ziemke, G., Hiebert, R., Weiser, S., Brinkmeyer, M., Fox, B., . . . Nordin, M. (2012). Implementation of a multidisciplinary program for active duty personnel seeking care for low back pain in a US Navy Medical Center: a feasibility study. *Military medicine*, 177(9), 1075-1080.
- 57. Weiser, S., Lis, A., Ziemke, G., Hiebert, R., Faulkner, D., Brennan, T., . . . Campello, M. (2018).
- Feasibility of Training Physical Therapists to Implement a Psychologically Informed Physical Therapy Program for Deployed U.S. Sailors and Marines with Musculoskeletal Injuries. *Mil Med*, 183(suppl 1), 503-509. doi:10.1093/milmed/usx229
- 58. Curran, G. M., Bauer, M., Mittman, B., Pyne, J. M., & Stetler, C. (2012). Effectiveness-implementation hybrid designs: combining elements of clinical effectiveness and implementation research to enhance public health impact. *Med Care*, 50(3), 217-226. doi:10.1097/MLR. 0b013e3182408812
- 59. Yates, S. L., Morley, S., Eccleston, C., & Williams, A. C. d. C. (2005). A scale for rating the quality of psychological trials for pain. *Pain*, 117(3), 314-325.
- 60. Tait, R. C., Pollard, C. A., Margolis, R. B., Duckro, P. N., & Krause, S. (1987). The Pain Disability Index: psychometric and validity data. Arch Phys Med Rehabil, 68(7), 438-441.
- 61. Sullivan, M. J., Bishop, S. R., & Pivik, J. (1995). The pain catastrophizing scale: Development and validation. . *Psychological Assessment*, 7, 524.
- 62. Waddell, G., Newton, M., Henderson, I., Somerville, D., & Main, C. J. (1993). A Fear-Avoidance Beliefs Questionnaire (FABQ) and the role of fear-avoidance beliefs in chronic low back pain and disability. *Pain*, 52. doi:10.1016/0304-3959(93)90127-b
- 63. George, S. Z., Fritz, J. M., & Childs, J. D. (2008). Investigation of elevated fear-avoidance beliefs for patients with low back pain: a secondary analysis involving patients enrolled in physical therapy clinical trials. *Journal of Orthopaedic & Sports Physical Therapy*, 38(2), 50-58.
- 64. Zigmond, A. S., & Snaith, R. P. (1983). The hospital anxiety and depression scale. *Acta Psychiatr Scand*, 67(6), 361-370. doi:10.1111/j.1600-0447.1983.tb09716.x
- 65. Herrmann, C. (1997). International experiences with the Hospital Anxiety and Depression Scale--a review of validation data and clinical results. *J Psychosom Res*, 42(1), 17-41. doi: 10.1016/s0022-3999(96)00216-4
- 66. Rusu, A. C., Santos, R., & Pincus, T. (2016). Pain-related distress and clinical depression in chronic pain: A comparison between two measures. *Scand J Pain*, 12, 62-67. doi:10.1016/j. sjpain.2016.04.001
- 67. Nicholas, M. K. (2007). The pain self-efficacy questionnaire: Taking pain into account. *Eur J Pain*, 11(2), 153-163. doi:10.1016/j.ejpain.2005.12.008

- 68. Cohen, M., Nicholas, M., & Blanch, A. (2000). Medical assessment and management of work-related low back or neck/arm pain. . *Journal of Occupational Health and Safety Australia and New Zealand*, 16, 307-318.
- 69. Adams, J. H., & Williams, A. C. (2003). What affects return to work for graduates of a pain management program with chronic upper limb pain? *J Occup Rehabil*, 13(2), 91-106. doi:10.1023/a:1022599731391
- 70. Coughlan, G. M., Ridout, K. L., Williams, A. C., & Richardson, P. H. (1995). Attrition from a pain management programme. *Br J Clin Psychol*, 34(3), 471-479. doi:10.1111/j.2044-8260.1995. tb01481.x
- 71. Beattie, P., Turner, C., Dowda, M., Michener, L., & Nelson, R. (2005). The MedRisk instrument for measuring patient satisfaction with physical therapy care: a psychometric analysis. *Journal of Orthopaedic & Sports Physical Therapy*, 35(1), 24-32.
- 72. Beattie, P. F., Pinto, M. B., Nelson, M. K., & Nelson, R. (2002). Patient satisfaction with outpatient physical therapy: instrument validation. *Phys Ther*, 82(6), 557-565.
- 73. Mannion, A. F., Porchet, F., Kleinstuck, F. S., Lattig, F., Jeszenszky, D., Bartanusz, V., . . . Grob, D. (2009). The quality of spine surgery from the patient's perspective. Part 1: the Core Outcome Measures Index in clinical practice. *Eur Spine J*, 18 Suppl 3, 367-373. doi:10.1007/s00586-009-0942-8
- 74. Radloff, L. S. (1977). The CES-D scale a self-report depression scale for research in the general population. *Applied Psychological Measurement*, 1, 385-401.
- 75. Radloff, L. S., & Locke, B. Z. (1986). The community mental health assessment survey and the CES-D scale. . *Community Surveys of Psychiatric Disorders*, 4, 177-188.
- 76. Lowe, B., Decker, O., Muller, S., Brahler, E., Schellberg, D., Herzog, W., & Herzberg, P. Y. (2008). Validation and standardization of the Generalized Anxiety Disorder Screener (GAD-7) in the general population. *Med Care*, 46(3), 266-274. doi:10.1097/MLR.0b013e318160d093
- 77. Bliese, P. D., Wright, K. M., Adler, A. B., Cabrera, O., Castro, C. A., & Hoge, C. W. (2008). Validating the primary care posttraumatic stress disorder screen and the posttraumatic stress disorder checklist with soldiers returning from combat. *J Consult Clin Psychol*, 76(2), 272-281. doi:10.1037/0022-006x.76.2.272
- 78. Weathers, F. W., Huska, J. A., & Keane, T. M. (1991). *PCL-M for DSM-IV*. Boston: National Center for PTSD Behavioral Science Division.
- 79. Dolbier, C. L., Webster, J. A., McCalister, K. T., Mallon, M. W., & Steinhardt, M. A. (2005). Reliability and validity of a single-item measure of job satisfaction. *Am J Health Promot*, 19(3), 194-198. doi:10.4278/0890-1171-19.3.194
- 80. Gade, P. A., Tiggle, R. B., & Schumm, W. R. (2003). The measurement and consequences of military organizational commitment in soldiers and spouses. *Military Psychology*, 14, 191-207.
- 81. Porter, L. W., & Smith, F. E. (1970). The etiology of organizational commitment: a longitudinal study of the initial stages of employee-organization reactions. University of California, Irvine.
- 82. Martin, T. N., & O'Laughlin, M. S. (1984). Predictors of organizational commitment: the study of parttime army reservists. . *Journal of Vocational Behavior*, 25, 270-283.
- 83. Rosen, L. N., & Martin, L. (1996). Childhood antecedents of psychological adaptation to military life. *Mil Med*, 161(11), 665-668.
- 84. Vogt, D. S., Proctor, S. P., King, D. W., King, L. A., & Vasterling, J. J. (2008). Validation of scales from the Deployment Risk and Resilience Inventory in a sample of Operation Iraqi Freedom veterans. *Assessment*, 15(4), 391-403. doi:10.1177/1073191108316030
- 85. Barell, V., Aharonson-Daniel, L., Fingerhut, L. A., Mackenzie, E. J., Ziv, A., Boyko, V., . . . Heruti, R. (2002). An introduction to the Barell body region by nature of injury diagnosis matrix. *I nj Prev*, 8(2), 91-96. doi:10.1136/jp.8.2.91
- 86. Keogh, A., Matthews, J., Segurado, R., & Hurley, D. A. (2018). Feasibility of Training Physical Therapists to Deliver the Theory-Based Self-Management of Osteoarthritis and Low Back Pain Through Activity and Skills (SOLAS) Intervention Within a Trial. *Phys Ther*, 98(2), 95-107. doi: 10.1093/ptj/pzx105

**ADSM - Active Duty Service Members** 

AHLTA - Armed forces Health Longitudinal Technology Application

CBT - Cognitive Behavioral Therapy.

CES-D - Center for Epidemiologic Studies Depression Scale

CID - Clinical Investigations Department at NMCP

COMI - Core Outcome Measures Index

CDMRP - Congressionally Directed Medical Research Programs

CRADA - Cooperative Research and Development Agreement

DRRI - Deployment Risk and Resilience Inventory-2

FAB - Fear avoidance beliefs

FABQ - Fear Avoidance Beliefs Questionnaire

GAD-7 - General Anxiety Disorder Screener

HADS - Hospital Anxiety and Depression Scale

ICD - International Classification of Diseases

IFC - Informed Consent Form

IRB - Institutional Review Board

LBP - Low Back Pain

MRPS - MedRisk Instrument for Measuring Patient Satisfaction

MSD - Musculoskeletal Disorders

NMCP - Navy Medical Center Portsmouth

NYU - New York University

PCL-M - PTSD Checklist Military Version

PCS - Pain Catastrophizing Scale

PDI - Pain Disability Index

PEB - Physical Evaluation Board

PHI - Personal Health Information

PI - Principle Investigator

PiPT - Psychologically-informed Physical Therapy

PSEQ - Pain Self-efficacy Questionnaire

PT - Physical Therapy

PTSD - Post-traumatic Stress Disorder

RA - Research Assistant

RCT - Randomized Controlled Trial

SOAP note - Subjective, Objective, Assessment, and Plan note